#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# **Clinical Study Protocol**

A Phase 3b Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Cystic Fibrosis Subjects Ages 6 Years and Older Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)

Vertex Study Number: VX20-445-119 EudraCT Number: 2020-001404-42

**Date of Protocol:** 26 June 2020 (Version 1.0)

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### 2 PROTOCOL SYNOPSIS

**Brief Title** 

Title A Phase 3b Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Cystic Fibrosis Subjects Ages 6 Years and Older Who Are Heterozygous

for the F508del Mutation and a Minimal Function Mutation (F/MF)

A Study Evaluating the Long-term Safety and Efficacy of

Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis (CF) Subjects 6 Years and Older and F/MF genotypes

Clinical Phase and Clinical Study Type

Phase 3b, safety, efficacy

#### **Objectives** Primary Objective

To evaluate the long-term safety and tolerability of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) in subjects with CF

#### **Secondary Objectives**

- To evaluate the efficacy of ELX/TEZ/IVA
- To evaluate the pharmacodynamics (PD) of ELX/TEZ/IVA

#### **Endpoints Primary Endpoint**

Safety and tolerability of ELX/TEZ/IVA based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry

#### **Secondary Endpoints**

- Absolute change in sweat chloride (SwCl) from baseline
- Absolute change in lung clearance index<sub>2.5</sub> (LCI<sub>2.5</sub>) from baseline

#### **Other Endpoints**

- Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline
- Absolute change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain score from baseline

#### **Number of Subjects**

Subjects who participated in the parent study (VX19-445-116) and meet the eligibility criteria may enroll. Approximately 108 subjects are expected to enroll in this extension study.

**Study Population** Male and female CF subjects who are 6 years of age or older who have F/MF genotypes.

#### Investigational Drug Active substance: ELX (VX-445)/TEZ (VX-661)/IVA (VX-770)

Activity: CFTR correctors (ELX and TEZ) and potentiator (IVA)

#### Strength and route of administration:

• 50-mg ELX/25-mg TEZ/37.5-mg IVA fixed-dose combination (FDC) tablets for oral administration

100-mg ELX/50-mg TEZ/75-mg IVA FDC tablets for oral administration

Active substance: IVA (VX-770)
Activity: CFTR potentiator

#### Strength and route of administration:

- 75-mg IVA tablets for oral administration
- 150-mg IVA tablets for oral administration

#### **Study Duration**

The total study duration is approximately 100 weeks (from the first dose of study drug in this study), including a Treatment Period of 96 weeks and a 4-week Safety Follow-up Visit.

#### Study Design

This is a Phase 3b, multicenter, open-label study for subjects who complete the parent study (VX19-445-116) and meet eligibility criteria. A schematic of the study design is shown in Figure 2-1.

Figure 2-1 VX20-445-119 Study Design



ELX: elexacaftor; IVA: ivacaftor, TEZ: tezacaftor

Note: Figure not drawn to scale.

Subjects will receive ELX/TEZ/IVA at the weight-appropriate dosage levels shown in Table 2-1 based on their weight at Day 1.

**Table 2-1** Treatment Period Dosages

| Subject Age | | | |
|-----------------|------------|------------|-------------|
| Weight | ELX Dosage | TEZ Dosage | IVA Dosage |
| ≥6 to <12 years | | | |
| <30 kg | 100 mg qd | 50 mg qd | 75 mg q12h |
| ≥30 kg | 200 mg qd | 100 mg qd | 150 mg q12h |
| ≥12 years | | | |
| All weights | 200 mg qd | 100 mg qd | 150 mg q12h |

ELX: elexacaftor; IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TEZ: tezacaftor

If a subject enters the current study weighing <30 kg and subsequently weighs  $\ge 30 \text{ kg}$  at 2 consecutive clinic visits (excluding unscheduled visits), the dose will be adjusted to the higher dose of ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for the remainder of the study, starting with the second visit where the subject's weight is  $\ge 30 \text{ kg}$ .

Subjects ≥12 years of age will receive a dose of ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h, starting from the first study visit at which the subject is ≥12 years old.

Assessments

**Safety:** AEs, clinical laboratory assessments, ECGs, vital signs, height, weight, pulse oximetry, physical examinations (PEs), and ophthalmologic examinations

Efficacy: Multiple-breath washout (MBW), spirometry, and CFQ-R

Pharmacodynamics (PD): SwCl

Other: blood samples for blood biomarker analysis

**Statistical Analyses** 

The primary objective of the study is the evaluation of the long-term safety and tolerability of ELX/TEZ/IVA in subjects with CF. The safety endpoints of long-term treatment include AEs, clinical laboratory values, ECGs, vital signs, and pulse oximetry from the first dose of study drug in the open label study, for subjects who have received at least 1 dose of study drug in the open label study. The safety analysis will be descriptive only, and in general will be performed for the pooled population.

The secondary objective of the study is the evaluation of long-term efficacy of ELX/TEZ/IVA, as assessed by SwCl, LCI<sub>2.5</sub>, spirometry, and CFQ-R. Methods of efficacy analyses will be similar as those used in parent studies

**Interim Analyses** 

Interim analyses may take place at any time at the discretion of the sponsor.

**DMC Reviews** 

A data monitoring committee (DMC) will conduct periodic safety review(s) of study data as outlined in the DMC charter.

### 3 SCHEDULE OF ASSESSMENTS

The schedule of assessments is in Table 3-1. All visits will be scheduled relative to the Day 1 Visit in this study.

Assessments may be performed in any order when more than 1 assessment is required at a particular time point, unless noted otherwise. All assessments should be performed before study drug dosing (Section 9.6), unless noted otherwise.

| | | | Treatment Per | iod | | | Safety | |
|---|---|---|---|---|---|---|---|---|
| Event/<br>Assessment <sup>a</sup> | Day<br>1 <sup>d</sup> | Weeks 4,<br>8, 16, 24<br>(± 5 Days) | Weeks 12, 20,<br>28, 32, 40, 44,<br>52, 56, 64, 68,<br>76, 80, 88, 92<br>(± 5 Days) | Weeks 36,<br>48, 60, 72,<br>84<br>(± 5 Days) | Week 96<br>(± 10 Days) | ETT Visit <sup>b</sup> | Follow-up Visit (28 ± 7 Days After Last Dose of Study Drug') | Comments |
| Clinic visit | X | X | | X | X | X | X | See Section 9.1.6 for use of remote measures in extenuating circumstances. |
| Telephone<br>contact | | | X | | | | | Assess subject's status, any AEs, concomitant medications, treatments, and procedures. |
| ICF and assent | X | | | | | | | |
| Safety and Efficac | y Assessi | ments | | | | | | |
| CFQ-R | X | X | | Weeks 48,<br>72 | X | | | Completed before the start of any other assessments (Section 11.2.4). |
| Ophthalmologic examination | | | | Week 48<br>(± 4 weeks) | X<br>(- 4 weeks) | X<br>(- 4 weeks) | X<br>(- 4 weeks) | Subjects will have an ophthalmologic examination at the completion of study participation (defined in Section 9.1.5). This examination should be completed at or up to 4 weeks before the relevant study visit (Section 11.4.6). |
| Height and<br>weight | X | X | | X | X | X | X | Measured with shoes off (Section 11.4.4). |
| Vital signs and pulse oximetry | X | X | | X | X | X | X | Performed after subject has been at rest for at least 5 minutes (Section 11.4.3). |
| Physical<br>examination (PE) | X | | | | X | X | | Symptom-directed PEs may be performed at any time if deemed necessary by the investigator (Section 11.4.3). |

a All assessments will be performed before dosing unless noted otherwise.

If the subject prematurely discontinues study drug treatment, an ETT Visit should be scheduled as soon as possible after the decision to discontinue treatment (Section 9.1.3).

<sup>&</sup>lt;sup>c</sup> The Safety Follow-up Visit is required for all subjects, unless otherwise specified. For subjects who complete an ETT Visit 3 weeks or later following the last dose of study drug, the ETT Visit will replace the Safety Follow-up Visit (Section 9.1.2).

The Day 1 Visit should be on the same day as the last scheduled visit of the parent study (Section 9.1.1). Subjects whose Day 1 Visit is NOT within 1 day of the last scheduled visit of the parent study will repeat all Day 1 assessments. Subjects whose Day 1 Visit is within 1 day of the last scheduled visit of the parent study will NOT have to repeat any Day 1 assessments that were specified to be performed at the last scheduled visit in the parent study.

| Table 3-1 | Table 3-1 Study VX20-445-119: Treatment Period and Safety Follow-up Visit | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Treatment Peri | od | | | Safety<br>Follow-up | |
| Event/<br>Assessment <sup>a</sup> | Day<br>1 <sup>d</sup> | Weeks 4,<br>8, 16, 24<br>(± 5 Days) | Weeks 12, 20,<br>28, 32, 40, 44,<br>52, 56, 64, 68,<br>76, 80, 88, 92<br>(± 5 Days) | Weeks 36,<br>48, 60, 72,<br>84<br>(± 5 Days) | Week 96<br>(± 10 Days) | ETT Visit <sup>b</sup> | Visit (28 ± 7 Days After Last Dose of Study Drug') | Comments |
| Standard 12-lead<br>ECG | X | Weeks 8,<br>16, 24 | | Weeks 48,<br>72 | X | X | X | Performed prior to any procedure that may affect heart rate (e.g., blood draws) and after subject has been at rest for at least 5 minutes (Section 11.4.5). |
| Sweat chloride | X | X | | Weeks 48,<br>72 | X | X | | Section 11.2.1 |
| Multiple-breath<br>washout | X | Х | | Weeks 48,<br>72 | Х | X | | Performed in multiple replicates,<br>pre-bronchodilator, before the AM dose, and<br>before spirometry assessment (Section 11.2.1). |
| Spirometry | X | X | | X | X | X | X | Performed pre-bronchodilator, before the AM dose, and at approximately the same time at each visit (Section 11.2.3). |
| Pregnancy test | Urine | Serum | Urine | Serum | Serum | Serum | Serum | For all female subjects at telephone contacts, a urine pregnancy test will be performed with a home kit provided by the study site. Results of the home pregnancy test will be reported to the site by telephone (Section 11.4.2). |
| Serum chemistry | X | X | | X | X | X | X | |
| Hematology | X | X | | X | X | X | X | |
| Coagulation | X | Week 24 | | Weeks 48,<br>72 | X | X | | Section 11.4.2 |
| Urinalysis | X | | | Week 48 | X | X | | |
| AEs and SAEs | | Continuo | us from signing of th | ne ICF through | completion of s | tudy participati | on | Section 13.1; Completion of study participation is defined in Section 9.1.5. |

| Table 3-1 | Study | VX20-445 | -119: Treatme | nt Period a | nd Safety l | Follow-up <b>V</b> | Visit | |
|---|---|---|---|---|---|---|---|---|
| | | | Treatment Peri | od | | | Safety | |
| Event/<br>Assessment <sup>a</sup> | Day<br>1 <sup>d</sup> | Weeks 4,<br>8, 16, 24<br>(± 5 Days) | Weeks 12, 20,<br>28, 32, 40, 44,<br>52, 56, 64, 68,<br>76, 80, 88, 92<br>(± 5 Days) | Weeks 36,<br>48, 60, 72,<br>84<br>(± 5 Days) | Week 96<br>(± 10 Days) | ETT Visit <sup>b</sup> | Follow-up Visit (28 ± 7 Days After Last Dose of Study Drug') | Comments |
| Medications review | | Continuous from signing of the ICF through completion of stu- | | | | | on | Completion of study participation is defined in Section 9.1.5. |
| Treatments and procedures review | | Continuous from signing of the ICF through completion of study participation | | | | | | |
| Biomarker Assessi | nent | | | | | | | |
| Blood biomarker collection | X | Week 24 | | Week 48 | X | X | | Section 11.3.1 |
| Study Drug Admir | istration | 1 | | , | - | | , | |
| ELX/TEZ/IVA | Day 1 through evening before Week 96 Visit | | | | | | | Subjects on study drug interruption from the parent study may NOT begin dosing until they meet the resumption criteria in Section 9.8. Refer to Section 9.6.1 for study drug administration details. |
| Study drug count | X | X | | X | X | X | | |

AE: adverse event; CFQ-R: Cystic Fibrosis Questionnaire-Revised; ELX: elexacaftor; ETT: early termination of treatment; ICF: informed consent form; IVA: ivacaftor; PE: physical examination: SAE: serious adverse event; TEZ: tezacaftor

# 4 TABLE OF CONTENTS

| I | | age | |
|---|------------|-----------------------------------------------------|----|
| 2 | Protoc | ol Synopsis | 2 |
| 3 | Schedu | lle of Assessments | 5 |
| 4 | Table ( | of Contents | 9 |
| | List of T | ables | 12 |
| | List of Fi | igures | 12 |
| | List of A | bbreviations | 13 |
| 5 | Introd | uction | 16 |
| | 5.1 Ba | ckground | 16 |
| | 5.2 Stu | ıdy Rationale | 16 |
| 6 | Study ( | Objectives | 16 |
| | 6.1 Pri | mary Objective | 16 |
| | 6.2 Sec | condary Objectives | 16 |
| 7 | Study I | Endpoints | 17 |
| | 7.1 Pri | mary Endpoint | 17 |
| | 7.2 Sec | condary Endpoints | 17 |
| | 7.3 Otl | her Endpoints | 17 |
| 8 | Study J | Population | 17 |
| | 8.1 Inc | clusion Criteria | 17 |
| | 8.2 Ex | clusion Criteria | 17 |
| 9 | Study J | Implementation | 18 |
| | 9.1 Stu | ıdy Design | 18 |
| | 9.1.1 | Treatment Period | 19 |
| | 9.1.2 | Follow-up | |
| | 9.1.3 | Early Termination of Treatment | 19 |
| | 9.1.4 | Lost to Follow-up | 20 |
| | 9.1.5 | Completion of Study Participation | |
| | 9.1.6 | Use of Remote Measures in Extenuating Circumstances | 20 |
| | | ethod of Assigning Subjects to Treatment Groups | |
| | 9.3 Ra | tionale for Study Elements | |
| | 9.3.1 | Study Design | |
| | 9.3.2 | Study Drug Dose and Duration | |
| | 9.3.3 | Rationale for Study Assessments | 21 |
| | | ıdy Restrictions | |
| | | or and Concomitant Medications | |
| | | lministration | |
| | 9.6.1 | Dosing | |
| | 9.6.2 | Missed Doses | |
| | | se Modification for Toxicity | |
| | | ndy Drug Interruption and Stopping Rules | |
| | 9.8.1 | Liver Function Tests | |
| | 9.8.2 | Rash | |
| | | moval of Subjects | |
| | 9.10 Re | placement of Subjects | 26 |

| <b>10</b> | Study Dru | ng Information and Management | 26 |
|---|---|---|---|
| | | ration and Dispensing | |
| | 10.2 Packa | ging and Labeling | 26 |
| | 10.3 Study | Drug Supply, Storage, and Handling | 26 |
| | - | Accountability | |
| | 10.5 Dispo | sal, Return, or Retention of Unused Drug | 27 |
| | | liance | |
| | | ng and Unblinding | |
| | | nts | |
| | 11.1 Subje | ct and Disease Characteristics | 28 |
| | 11.2 Effica | cy and Pharmacodynamics | 28 |
| | | weat Chloride | |
| | 11.2.2 N | Aultiple-breath Washout | 28 |
| | 11.2.3 S | pirometry | 28 |
| | 11.2.4 | Cystic Fibrosis Questionnaire-Revised | 29 |
| | 11.3 Other | Assessments | 30 |
| | 11.3.1 E | Blood Biomarkers | 30 |
| | 11.4 Safety | <sup>7</sup> | 30 |
| | 11.4.1 A | Adverse Events | 30 |
| | 11.4.2 | Clinical Laboratory Assessments | 30 |
| | 11.4.3 F | Physical Examinations and Vital Signs | 32 |
| | 11.4.4 H | leight and Weight | 32 |
| | 11.4.5 E | Electrocardiograms | 32 |
| | 11.4.6 | Ophthalmologic Examination | 32 |
| | 11.4.7 | Contraception and Pregnancy | 33 |
| | 11.4.7. | Contraception | 33 |
| | 11.4.7.2 | Pregnancy | 34 |
| 12 | Statistical | Analysis | 35 |
| | 12.1 Samp | le Size | 35 |
| | 12.2 Analy | sis Sets | 35 |
| | 12.3 Statist | ical Analysis | 35 |
| | 12.3.1 | General Considerations | 35 |
| | 12.3.2 E | Background Characteristics | 36 |
| | 12.3.2. | | |
| | 12.3.2.2 | 2 Demographics and Baseline Characteristics | 36 |
| | 12.3.2.3 | Prior and Concomitant Medications | 37 |
| | 12.3.2.4 | Study Drug Exposure and Compliance | 37 |
| | 12.3.2.5 | | 37 |
| | 12.3.3 E | Efficacy Analysis | |
| | 12.3.3. | Analysis of Primary Efficacy and Pharmacodynamic Endpoints | 38 |
| | 12.3.3.2 | 2 Analysis of Secondary Efficacy and Pharmacodynamic Endpoints | 38 |
| | 12.3.3.3 | • | |
| | 12.3.3.4 | | |
| | 12.3.4 S | afety Analysis | |
| | 12.3.4.1 | | |
| | 12.3.4.2 | 2 Clinical Laboratory Assessments | 40 |

| | 12.3.4.3 | Electrocardiogram | 40 |
|---|---|---|---|
| | 12.3.4.4 | Vital Signs | 40 |
| | 12.3.4.5 | Pulse Oximetry | 40 |
| | 12.3.4.6 | Physical Examination | |
| | 12.3.4.7 | Other Safety Analyses | |
| | 12.4 Interim | Analysis | |
| | 12.5 Data M | onitoring Committee Analysis | 41 |
| 13 | | , Ethical, Regulatory, and Administrative Considerations | |
| | | E Event and Serious Adverse Event Documentation, Severity Grading, and | |
| | | ng | 41 |
| | | verse Events | |
| | 13.1.1.1 | Definition of an Adverse Event | |
| | 13.1.1.2 | Clinically Significant Assessments | |
| | 13.1.1.3 | Documentation of Adverse Events | |
| | 13.1.1.4 | Adverse Event Severity | 42 |
| | 13.1.1.5 | Adverse Event Causality | |
| | 13.1.1.6 | Study Drug Action Taken | |
| | 13.1.1.7 | Adverse Event Outcome | |
| | 13.1.1.8 | Treatment Given | 44 |
| | 13.1.2 Sea | rious Adverse Events | 44 |
| | 13.1.2.1 | Definition of a Serious Adverse Event. | 44 |
| | 13.1.2.2 | Reporting and Documentation of Serious Adverse Events | 45 |
| | 13.1.2.3 | | |
| | | strative Requirements | |
| | | oduct Complaints | |
| | | nical Considerations | |
| | | bject Information and Informed Consent | |
| | | Vestigator Compliance | |
| | | cess to Records. | |
| | 13.2.6 Su | bject Privacy | 47 |
| | | cord Retention | |
| | 13.2.8 Stu | ady Termination | 47 |
| | 13.2.9 En | d of Study | 48 |
| | | uality Assurance | |
| | | ring | |
| | | nic Data Capture | |
| | | entiality and Disclosure | |
| | | tions and Clinical Study Report | |
| | | blication of Study Results | |
| | | inical Study Report | |
| 14 | | | |
| | | gnature Pages | |
| | • | r Signature Page | |
| | | gator Signature Page | |

# **List of Tables**

| Treatment Period Dosages | 3 |
|---|---|
| Study VX20-445-119: Treatment Period and Safety Follow-up Visit | 6 |
| Treatment Period Dosages | 18 |
| Prohibited Medications | 22 |
| Study Drug Administration | 23 |
| Study Drug: Dosing Form/Route/Strength | 27 |
| Safety Laboratory Test Panels | 31 |
| Acceptable Methods of Contraception | 34 |
| Grading of AE Severity | |
| Classifications for AE Causality | 43 |
| Classifications for Study Drug Action Taken With Regard to an AE | 43 |
| Classifications for Outcome of an AE | |
| res | |
| VX20-445-119 Study Design | 3 |
| VX20-445-119 Study Design | 18 |
| | Treatment Period Dosages Prohibited Medications Study Drug Administration Study Drug: Dosing Form/Route/Strength Safety Laboratory Test Panels Acceptable Methods of Contraception. Grading of AE Severity Classifications for AE Causality Classifications for Study Drug Action Taken With Regard to an AE Classifications for Outcome of an AE VX20-445-119 Study Design |

# **List of Abbreviations**

| ADL activities of daily living AES adverse events ALT alanine transaminase AST aspartate transaminase β beta, apparent elimination rate constant BMI body mass index CD compact disc CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electrocardiogram EDC electroic data capture EENT eyes, cars, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEFQ-150-75% forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative GPP3 Good Publishing Practices | Abbreviation | Definition |
|---|---|---|
| ALT alanine transaminase AST aspartate transaminase β beta, apparent elimination rate constant BMI body mass index CD compact dise CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electroic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union FMF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEF25%-75% forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | | |
| AST aspartate transaminase β beta, apparent elimination rate constant BMI body mass index CD compact disc CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | AEs | adverse events |
| β beta, apparent elimination rate constant BMI body mass index CD compact disc CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FEF25%-75% forced expiratory flow, midexpiratory phase | ALT | alanine transaminase |
| BMI body mass index CD compact disc CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, cars, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEE25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | AST | aspartate transaminase |
| CD compact disc CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | β | beta, apparent elimination rate constant |
| CF Cystic Fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG clectrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEC forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | BMI | body mass index |
| CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CD | compact disc |
| CFTR CF transmembrane conductance regulator gene CI confidence interval COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CF | Cystic Fibrosis |
| CI confidence interval coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT cyes, cars, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CFQ-R | Cystic Fibrosis Questionnaire-Revised |
| COVID-19 coronavirus disease CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CFTR | CF transmembrane conductance regulator gene |
| CRF clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, cars, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CI | confidence interval |
| CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | COVID-19 | coronavirus disease |
| CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CRF | case report form |
| CYP cytochrome P450 DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CSR | clinical study report |
| DMC data monitoring committee ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CTCAE | Common Terminology Criteria for Adverse Events |
| ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | CYP | cytochrome P450 |
| EDC electronic data capture EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | DMC | data monitoring committee |
| EENT eyes, ears, nose, and throat ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | ECG | electrocardiogram |
| ELX elexacaftor ETT Early Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | EDC | electronic data capture |
| ETT Eurly Termination of Treatment EU European Union F/MF F508del Mutation and a Minimal Function Mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | EENT | eyes, ears, nose, and throat |
| EU European Union F/MF F508del Mutation and a Minimal Function Mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | ELX | elexacaftor |
| F/MF F508del Mutation and a Minimal Function Mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | ETT | Early Termination of Treatment |
| F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | EU | European Union |
| codon corresponding to position 508 of the wild-type protein FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | F/MF | F508del Mutation and a Minimal Function Mutation |
| FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | F508del | |
| FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | FDA | Food and Drug Administration |
| FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | FDC | fixed-dose combination |
| FSH follicle-stimulating hormone FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | FEF25%-75% | forced expiratory flow, midexpiratory phase |
| FVC Forced vital capacity GCP Good Clinical Practice GLI Global Lung Function Initiative | FEV <sub>1</sub> | forced expiratory volume in 1 second |
| GCP Good Clinical Practice GLI Global Lung Function Initiative | FSH | follicle-stimulating hormone |
| GLI Global Lung Function Initiative | FVC | Forced vital capacity |
| 3 | GCP | Good Clinical Practice |
| GPP3 Good Publishing Practices | GLI | Global Lung Function Initiative |
| | GPP3 | Good Publishing Practices |

| Abbreviation | Definition |
|---|---|
| GPS | Global Patient Safety |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | heart rate |
| ICF | informed consent form |
| ICH | International Council for Harmonization |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | independent ethics committee |
| IMP | investigational medicinal product |
| IPD | important protocol deviation |
| IRB | institutional review board |
| IVA | ivacaftor |
| IWRS | interactive web response system |
| LCI | lung clearance index |
| LCI <sub>2.5</sub> | number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value |
| LS | least squares |
| LUM | lumacaftor |
| max | maximum value |
| MBW | Multiple-breath washout |
| MedDRA | Medical Dictionary for Regulatory Activities |
| min | minimum value |
| MMRM | mixed-effects model for repeated measures |
| N | total sample size |
| OATP1B1 | organic anion transporting polypeptide 1B1 |
| OATP1B3 | organic anion transporting polypeptide 1B3 |
| OL-FAS | Open-label Full Analysis Set |
| OL-SS | Open-label Safety Set |
| PC | publication committee |
| PD | pharmacodynamics |
| PEs | physical examinations |
| P-gp | P-glycoprotein |
| PIs | principal investigators |
| ppFEV <sub>1</sub> | percent predicted forced expiratory volume in 1 second |
| PR | PR interval, segment |
| PT | Preferred Term |
| q12h | every 12 hours |

| Abbreviation | Definition |
|---|---|
| qd | once daily |
| QRS | the portion of an ECG comprising the Q, R, and S waves, together representing ventricular depolarization |
| QT | QT interval |
| QTcF | QT interval corrected by Fridericia's formula |
| RNA | ribonucleic acid |
| RR | interval from the onset of 1 QRS complex to the next; use R-R if using with "intervals", i.e., "R-R interval" |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SC | steering committee |
| SD | standard deviation |
| SET | Study Execution Team |
| SI | SI units (International System of Units) |
| SOC | System Organ Class |
| SUSARs | serious adverse reactions |
| SwCl | sweat chloride |
| TE | Treatment-emergent |
| TEAEs | treatment-emergent adverse events |
| TEZ | tezacaftor |
| ULN | upper limit of normal |
| US | United States |
| USA | United States of America |
| VAS | visual analog scale |

#### 5 INTRODUCTION

### 5.1 Background

Cystic fibrosis (CF) is an autosomal recessive genetic disease with serious morbidities and frequent premature mortality. CF affects more than 70,000 individuals worldwide<sup>1</sup> (approximately 31,000 in the US<sup>2</sup> and 48,000 in the EU<sup>3</sup>).

CF is caused by decreased quantity and/or function of the CFTR protein due to mutations in the *CFTR* gene.<sup>4</sup> CFTR is a channel that regulates the flow of chloride and other anions across epithelia in multiple organs and tissues, including the lungs, pancreas and other gastrointestinal organs, and sweat glands.<sup>5</sup> Despite progress in the treatment of CF with antibiotics and mucolytics, the current median age at death among people with CF is approximately 30 years, and the predicted median age of survival is approximately 47 years.<sup>2, 3</sup> More effective treatments are needed for CF.

The most common disease-causing mutation is F508del: approximately 84.7% of people with CF in the US and 81.1% in Europe have at least one F508del allele.<sup>2, 3</sup>

At present CF does not have a cure. CFTR modulators (i.e., correctors and potentiators) represent a major advancement in the treatment of CF because they are systemic therapies that target the underlying cause of the disease and have been shown to improve CF survival by modifying the course of disease. <sup>6,7</sup> The clinical testing and regulatory approval of CFTR modulators in certain countries for the treatment of people with CF caused by specific *CFTR* genotypes has established the therapeutic value of specific regimens developed by Vertex. These treatment regimens include ivacaftor (IVA) monotherapy (Kalydeco<sup>TM</sup>), lumacaftor (LUM)/IVA dual combination therapy (Orkambi<sup>TM</sup>), tezacaftor (TEZ)/IVA dual combination therapy (Symdeko<sup>TM</sup>, Symkevi<sup>TM</sup>) and elexacaftor (ELX)/TEZ/IVA triple combination therapy.

The ELX/TEZ/IVA regimen is the first medicine to demonstrate clinical benefit in patients with a single *F508del* allele, regardless of the mutation of the second allele. A pivotal Phase 3 program in CF subjects 12 years of age or older demonstrated that ELX/TEZ/IVA provides substantial improvements in lung function, CFTR function, and nutritional status, and was generally safe and well tolerated with a low rate of treatment discontinuation.

### 5.2 Study Rationale

This study will provide data on the long-term safety and efficacy of ELX/TEZ/IVA in subjects with CF who are 6 years of age and older.

#### 6 STUDY OBJECTIVES

### 6.1 Primary Objective

To evaluate the long-term safety and tolerability of ELX/TEZ/IVA in subjects with CF

### 6.2 Secondary Objectives

- To evaluate the efficacy of ELX/TEZ/IVA
- To evaluate the pharmacodynamics (PD) of ELX/TEZ/IVA

### 7 STUDY ENDPOINTS

### 7.1 Primary Endpoint

Safety and tolerability of ELX/TEZ/IVA based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry

### 7.2 Secondary Endpoints

- Absolute change in sweat chloride (SwCl) from baseline
- Absolute change in lung clearance index2.5 (LCI2.5) from baseline

### 7.3 Other Endpoints

- Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline
- Absolute change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain score from baseline

#### 8 STUDY POPULATION

Eligibility will be reviewed and documented by an appropriately qualified member of the investigator's team before subjects are enrolled.

Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be eligible. In the criteria below, "parent study" is defined as VX19-445-116.

#### 8.1 Inclusion Criteria

- 1. Subject (or his or her legally appointed and authorized representative) will sign and date an informed consent form (ICF) and, when appropriate, an assent form.
- 2. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
- 3. Did not withdraw consent from the parent study.
- 4. Meets at least 1 of the following criteria:
  - Completed study drug treatment in the parent study.
  - Had study drug interruption(s) in the parent study, but did not permanently discontinue study drug, and completed study visits up to the last scheduled visit of the Treatment Period of the parent study.
- 5. Willing to remain on a stable CF treatment regimen (as defined in Section 9.5) through completion of study participation.

#### 8.2 Exclusion Criteria

- 1. History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
- 2. History of drug intolerance in the parent study that would pose an additional risk to the subject in the opinion of the investigator (e.g., subjects with a history of allergy or hypersensitivity to the study drug).

- 3. Pregnant and breast-feeding females. Female subjects must have a negative pregnancy test at the Day 1 Visit before receiving the first dose of study drug.
- 4. Current participation in an investigational drug trial other than the parent study. Participation in a noninterventional study (including observational studies, registry studies, and studies requiring blood collections without administration of study drug) and screening for another Vertex study is permitted.

#### 9 STUDY IMPLEMENTATION

# 9.1 Study Design

This is a Phase 3b, multicenter, open-label study for subjects who complete the parent study (VX19-445-116) and meet eligibility criteria. A schematic of the study design is shown in Figure 9-1.

Study visits and assessments to be conducted are shown in Table 3-1. All visits will occur within the windows specified.

Figure 9-1 VX20-445-119 Study Design



ELX: elexacaftor; IVA: ivacaftor, TEZ: tezacaftor

Note: Figure not drawn to scale.

Subjects will receive ELX/TEZ/IVA at the weight-appropriate dosage levels shown in Table 9-1 based on their weight at Day 1.

**Table 9-1** Treatment Period Dosages

| Subject Age<br>Weight | ELX Dosage | TEZ Dosage | IVA Dosage |
|---|---|---|---|
| ≥6 to <12 years | | | |
| <30 kg | $100~\mathrm{mg}~\mathrm{qd}$ | $50 \mathrm{\ mg\ qd}$ | 75 mg q12h |
| ≥30 kg | $200~\mathrm{mg}~\mathrm{qd}$ | $100 \mathrm{\ mg\ qd}$ | $150 \ \mathrm{mg} \ \mathrm{q}12\mathrm{h}$ |
| ≥12 years | | | |
| All weights | $200~\mathrm{mg}~\mathrm{qd}$ | $100 \mathrm{\ mg\ qd}$ | 150 mg q12h |

ELX: elexacaftor; IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TEZ: tezacaftor

Note: Study drug administration is described in Section 9.6.

If a subject enters the current study weighing <30 kg and subsequently weighs  $\ge 30 \text{ kg}$  at 2 consecutive clinic visits (excluding unscheduled visits), the dose will be adjusted to the higher dose of ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for the remainder of the study, starting with the second visit where subject's weight is  $\ge 30 \text{ kg}$ .

Subjects ≥12 years of age will receive a dose of ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h, starting from the first study visit at which the subject is ≥12 years old.

#### 9.1.1 Treatment Period

Treatment Period assessments are listed in Table 3-1.

Subjects will receive the first dose of study drug on Day 1 after obtaining informed consent (and assent, when applicable) and confirming eligibility. Subjects who enroll in this study on a study drug interruption will NOT receive the first dose of study drug until they meet the resumption criteria in Section 9.8; before receiving study drug, subjects will repeat all Day 1 assessments.

Study drug administration details are provided in Section 9.6.

Subjects whose Day 1 Visit is NOT within 1 day of the last scheduled visit of the parent study will repeat all Day 1 assessments.

Subjects whose Day 1 Visit is within 1 day of the last scheduled visit of the parent study will NOT have to repeat any Day 1 assessments that were specified to be performed at the last scheduled visit in the parent study.

#### 9.1.2 Follow-up

The Safety Follow-up Visit is scheduled to occur  $28 (\pm 7)$  days after the last dose of study drug. The Safety Follow-up Visit assessments are listed in Table 3-1.

The Safety Follow-up Visit is required for all subjects. However, subjects who transition within 28 days of the last dose of study drug to either:

- a commercially available Vertex CFTR modulator regimen
- managed access program-supplied Vertex CFTR modulator regimen
- or, to another qualified Vertex study

will complete the Week 96 Visit (or the Early Termination of Treatment [ETT] Visit, if the transition occurs before the Week 96 Visit). In these cases, the Week 96 Visit (or the ETT Visit) will replace the Safety Follow-up Visit.

For subjects who complete an ETT Visit 3 weeks or later following the last dose of study drug, the ETT Visit will replace the Safety Follow-up Visit (Section 9.1.3).

#### 9.1.3 Early Termination of Treatment

If a subject prematurely discontinues study drug treatment, an ETT Visit should be scheduled as soon as possible after the decision to discontinue treatment.

If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit.

If a subject withdraws from the study and also withdraws consent or assent, no further assessments will be performed. Vertex may retain and continue to use any data and samples collected before such withdrawal of consent or assent.

### 9.1.4 Lost to Follow-up

A subject will be considered lost to follow-up if both of the following occur:

- The subject misses 2 consecutive study visits (telephone contact and/or clinic visit) and is subsequently unable to be contacted by telephone (3 documented attempts by telephone within 2 weeks following the second missed visit)
- The subject does not respond within 2 weeks to a registered letter sent after the 3 attempted telephone contacts.

### 9.1.5 Completion of Study Participation

Completion of study participation for each individual subject is defined as: the Safety Follow-up Visit; or, in situations in which the ETT Visit or the Week 96 Visit replaces the Safety Follow-up Visit (Section 9.1.2), the ETT Visit or the Week 96 Visit.

If subjects withdraw consent or assent, completion of study participation is defined as date of withdrawal of consent or assent, whichever is earlier (Section 9.9).

If subjects are lost to follow-up (Section 9.1.4), the date of completion of study participation will be defined as the date of last contact.

The end of study is defined in Section 13.2.9.

### 9.1.6 Use of Remote Measures in Extenuating Circumstances

Study visits should be performed in the clinic as specified in Table 3-1, if at all possible. However, under extenuating circumstances, remote measures may be implemented (e.g., if a subject is unable to travel to the study site due to safety concerns and/or local restrictions related to COVID-19 or other emerging events). The decision whether to conduct study visits remotely or in clinic will be at the discretion of the investigator; if the investigator determines that study visits will be conducted remotely, the medical monitor should be notified. The Day 1 Visit must be performed in the clinic.

Whenever local regulations or site practice do not allow remote measures, visits will be conducted at the site.

The following remote measures may be implemented. Additional details can be found in the Study Reference Manual.

- Consent or reconsent may be obtained remotely in writing (or verbally, with follow-up written confirmation), as allowed by local regulations.
- Study drug may be shipped directly from the site to the subject, as applicable and as allowed by local regulations.
- Study visits (except Day 1) may be conducted as in-home visits by qualified personnel.
- Study assessments may be performed or overseen by qualified personnel conducting the in-home visits, except for multiple-breath washout (MBW) assessments.

• Remote monitoring visits may be implemented as applicable (including remote source data verification) and as allowed per local regulations.

## 9.2 Method of Assigning Subjects to Treatment Groups

This is an open-label study.

### 9.3 Rationale for Study Elements

### 9.3.1 Study Design

This Phase 3b study will enroll subjects who completed the last Treatment Period visit in the parent study of ELX/TEZ/IVA and meet eligibility criteria. Results from this study will provide information on the long-term safety and efficacy of ELX/TEZ/IVA in subjects with CF who are 6 years of age and older.

### 9.3.2 Study Drug Dose and Duration

To evaluate safety, tolerability, and efficacy, the study drug doses evaluated are the same as the doses evaluated in the parent study. Subjects will receive a study drug dose appropriate for their age and weight (as applicable), as described in Section 9.1.

The overall treatment duration will be 96 weeks, which is considered sufficient for evaluating the long-term safety and efficacy of ELX/TEZ/IVA treatment in individual subjects at the current stage of clinical development.

### 9.3.3 Rationale for Study Assessments

Most of the safety, efficacy, and PD assessments are standard parameters for clinical studies in drug development and are generally recognized as reliable, accurate, and relevant to the study of subjects with CF. Ophthalmologic examinations are recommended for monitoring of pediatric patients treated with IVA-containing drug regimens, and have been added to the standard safety assessments.

LCI is a measure of ventilation inhomogeneity assessed by MBW that is based on tidal breathing techniques that have been evaluated in patients as young as infants.<sup>8,9</sup> Studies have shown that LCI correlates with  $FEV_1$  in its ability to measure airway disease and can detect lung disease at an earlier stage than spirometry.<sup>10,11</sup>

### 9.4 Study Restrictions

Table 9-2 lists prohibited medications. A non-exhaustive list of study prohibitions and cautions for medication will be provided in the Study Reference Manual. Guidance for concomitant medications is provided in Section 9.5.

| | Timing of Restriction | | |
|---|---|---|---|
| Medication | Start of<br>Restriction | End of<br>Restriction | –<br>Rationale |
| Moderate and strong CYP3A inducers | None allowed<br>within 14 days<br>before the first<br>dose of the study<br>drug on Day 1 | None allowed<br>through<br>completion of<br>study<br>participation | ELX, TEZ, and IVA are metabolized extensively via CYP3A4. Therefore, use of moderate and strong inducers of CYP3A and |
| Moderate and strong<br>CYP3A inhibitors<br>(except<br>ciprofloxacin) <sup>a</sup> | None allowed<br>within 14 days<br>before the first<br>dose of the study<br>drug on Day 1 | None allowed<br>through<br>completion of<br>study<br>participation | moderate and strong inhibitors of CYP3A, which have the potential to alter the exposur of ELX, TEZ, or IVA, are prohibited. |
| CFTR modulators<br>(investigational or<br>approved), except for<br>study drugs in the<br>parent study and this<br>study | None allowed<br>within 28 days or<br>5 terminal half-<br>lives (whichever is<br>longer) before the<br>first dose of the<br>study drug on<br>Day 1 | None allowed<br>until after the<br>last dose of<br>study drug | These agents may confound the results of this study. |

**Table 9-2** Prohibited Medications

CYP: cytochrome P450; ELX: elexacaftor; IVA: ivacaftor; TEZ: tezacaftor

#### 9.5 Prior and Concomitant Medications

Information regarding prior and concomitant medications, including CF medications, other medications, and herbal and naturopathic remedies, will be collected in each subject's source documentation for medications taken within the 56 days before the first dose of study drug in this study through completion of study participation, as defined in Section 9.1.5.

- Subjects should remain on a stable treatment regimen for their CF through completion of study participation. Stable treatment regimen is defined as the current treatment regimen for CF that subjects have been following for at least 28 days before Day 1. Subjects should not initiate long-term treatment with new medication from 28 days before the Day 1 Visit through completion of study participation. Guidelines for stable treatment regimens for CF are as follows:
  - o Subjects who are taking inhaled tobramycin or other chronically inhaled antibiotics should remain on that regimen throughout the study.
  - o Subjects who cycle onto and off of an inhaled antibiotic should continue on their prior schedule.
  - o Subjects who alternate between 2 different inhaled antibiotics should remain on the same cycling schedule during the study.
- Subjects may receive doses of prednisone or prednisolone of up to 10 mg/day chronically, or up to 60 mg daily for up to 5 days.

Ciprofloxacin is not a moderate CYP3A inhibitor on the basis of results of a drug-drug interaction study conducted with IVA, a sensitive CYP3A substrate (Kalydeco [ivacaftor] US Package Insert).

- ELX may inhibit OATP1B1 and OATP1B3, which may increase the exposure of medicinal products that are substrates for these transporters. Substrates such as statins, glyburide, nateglinide, and repaglinide should be used with caution.
- IVA is a weak inhibitor of P-glycoprotein (P-gp). Administration of IVA may increase systemic exposure of medicinal products that are sensitive substrates of P-gp, which may increase or prolong their therapeutic effect and adverse reactions. Digoxin or other substrates of P-gp with a narrow therapeutic index, such as cyclosporine, everolimus, sirolimus, and tacrolimus, should be used with caution and appropriate monitoring.
- IVA may inhibit CYP2C9; therefore, during coadministration with warfarin, additional monitoring of the international normalized ratio is recommended. Other medicinal products that are CYP2C9 substrates for which exposure may be increased include glimepiride and glipizide; these should be used with caution.
- Information about bronchodilator use during the study will be collected and documented. Subjects who are using a bronchodilator should have their spirometry assessments performed according to the guidelines provided in Section 11.2.3.

#### 9.6 Administration

### **9.6.1 Dosing**

Study drug will be administered orally as shown in Table 9-3. Additional information is provided in the Pharmacy Manual.

**Table 9-3 Study Drug Administration** 

| Subject Age<br>Weight | Tablet Strength | Time | Number of Tablets Taken |
|---|---|---|---|
| ≥6 to <12 years | 50-mg ELX/25-mg TEZ/37.5-mg IVA | AM | 2 tablets |
| <30 kg | 75-mg IVA | PM | 1 tablet |
| ≥6 to <12 years | 100-mg ELX/50-mg TEZ/75-mg IVA | AM | 2 tablets |
| ≥30 kg | 150-mg IVA | PM | 1 tablet |
| ≥12 years | 100-mg ELX/50-mg TEZ/75-mg IVA | AM | 2 tablets |
| All weights | 150-mg IVA | PM | 1 tablet |

ELX: elexacaftor; IVA: ivacaftor; TEZ: tezacaftor

Study drug should be administered with a fat-containing meal or snack, such as a standard "CF" meal or snack or a standard meal according to the following guidelines:

- 1. It is recommended that the dose be taken within 30 minutes of the start of the meal or snack.
- 2. Study drug will be administered as 2 ELX/TEZ/IVA FDC tablets in the morning (see Table 9-3 for details) and as 1 IVA tablet in the evening. All doses of study drug (morning and evening, as applicable) should be administered at approximately every 12 hours (± 2 hours) on each dosing occasion (e.g., if the morning doses of study drug are administered at 08:00 hour on Day 1, all subsequent morning doses should be administered between 06:00 hour and 10:00 hour).

- 3. On days of scheduled visits, the morning dose of ELX/TEZ/IVA will be administered at the site after predose assessments have been completed. The meal or snack will be provided by the site for the morning dose of ELX/TEZ/IVA.
- 4. Subjects will be instructed to bring all used and unused materials associated with the study drug to the site; study drug will be dispensed at each visit, as appropriate.

#### 9.6.2 Missed Doses

If 6 hours or less have passed since the missed morning or evening dose, the subject should take the missed dose as soon as possible and continue on the original schedule.

**Morning dose:** If more than 6 hours have passed since the missed **morning** dose, the subject should take the missed dose as soon as possible and should not take the evening dose.

**Evening dose:** If more than 6 hours have passed since the missed **evening** dose, the subject should not take the missed dose. The next scheduled morning dose should be taken at the usual time.

Morning and evening doses should not be taken at the same time.

# 9.7 Dose Modification for Toxicity

No dose modifications for toxicity are allowed. If any unacceptable toxicity arises, individual subjects will discontinue dosing.

### 9.8 Study Drug Interruption and Stopping Rules

In subjects who have interrupted study drug for >72 hours for any reason, the investigator should resume study drug only after a thorough investigation of the cause for interruption. The investigator will evaluate the subject's clinical stability and should consider resumption of study drug only after the subject is clinically stable and there is no comorbidity or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.

The medical monitor should be notified of an interruption of study drug that lasts >72 hours for any reason and of the resumption of study drug after such interruption. In subjects for whom study drug was previously interrupted, the medical monitor should be notified of any plan to discontinue study drug, before the discontinuation has occurred, if possible.

#### 9.8.1 Liver Function Tests

The central laboratory will notify the medical monitor of alanine transaminase (ALT) or aspartate transaminase (AST) >3 × upper limit of normal (ULN) and total bilirubin >2 × ULN that are derived from centrally submitted samples.

Subjects with new treatment-emergent ALT or AST elevations of  $>3 \times ULN$ , with or without total bilirubin  $>2 \times ULN$ , must be followed closely, including confirmatory testing performed by the central laboratory within 48 to 72 hours of the initial finding and subsequent close monitoring of ALT, AST, and bilirubin levels, as clinically indicated.

If a subject cannot return to the site for confirmatory testing, a local laboratory may be used. Local laboratory results must be reported immediately to the medical monitor, and the subject must have the tests repeated and sent to the central laboratory as soon as possible (ideally within 48 to 72 hours).

Study drug administration <u>must be interrupted</u> immediately (prior to confirmatory testing) if any of the following criteria are met:

- ALT or AST >8 × ULN
- ALT or AST >5 × ULN for more than 2 weeks
- ALT or AST >3 × ULN, in association with total bilirubin >2 × ULN and/or clinical jaundice

A thorough investigation of potential causes should be conducted, and the subject should be followed closely for clinical progression.

Subjects who enroll in this study on a drug interruption because of transaminase elevations in a parent study may NOT receive the first dose of study drug until transaminases return to baseline values or  $\leq 2 \times \text{ULN}$ , whichever is higher.

Study drug administration **must be discontinued** if the following criteria are met:

• Subsequent ALT or AST values confirm the initial elevation that satisfied the interruption rule (above), and no convincing alternative etiology (e.g., acetaminophen use, viral hepatitis, alcohol ingestion) is identified, regardless of whether transaminase levels have improved

All subjects in whom treatment is discontinued for elevated transaminases (and bilirubin, as applicable) should have these levels monitored closely until levels normalize or return to baseline.

If an alternative, reversible cause of transaminase elevation with or without increased bilirubin or clinical jaundice has been identified, study drug administration may be resumed once transaminase levels return to baseline or are ≤2 × ULN, whichever is higher. Regardless of the duration of interruption, the medical monitor should be notified before resumption of study drug. Upon resumption of study drug, transaminases and bilirubin should be assessed weekly for 4 weeks. If a protocol-defined transaminase elevation interruption threshold recurs within 4 weeks of rechallenge with the study drug (with confirmation of the initial elevation by repeat testing within 48 to 72 hours), then the study drug must be permanently discontinued, regardless of the presumed etiology.

#### 9.8.2 Rash

Individuals who develop a generalized rash will be monitored closely. Study drug dosing should be interrupted if a subject develops a generalized rash of Grade 3 or higher (Section 13.1.1.4), or a rash that is considered a serious adverse event (SAE). The investigator will notify the medical monitor of any rash that results in interruption of study drug, is Grade 3 or higher, or is an SAE. Investigators should consider additional evaluation including laboratory testing (e.g., complete blood count with differential, liver function tests), photographs of the rash, and dermatology consultation. The investigator may consider resumption of study drug if considered clinically appropriate.

### 9.9 Removal of Subjects

Subjects may withdraw from the study at any time at their own request or the request of the subject's parent or legal guardian. Subjects may be withdrawn at any time at the discretion of the investigator or Vertex for safety, behavior, noncompliance (study drug dosing or study

procedures), or administrative reasons. A subject who withdraws from study drug treatment will continue to be followed unless the subject withdraws consent.

In addition, a subject must be discontinued from study drug treatment if the subject meets any of the following criteria:

- Meets any of the stopping (discontinuation) criteria (Section 9.8)
- Becomes pregnant (Section 11.4.7.2)

If a subject does not return for a scheduled visit, reasonable effort will be made to contact the subject. In any circumstance, reasonable effort will be made to document subject outcome. The investigator will inquire about the reason for withdrawal, request that the subject return all unused investigational product(s), request that the subject return for a Safety Follow-up Visit, if applicable (see Section 9.1.3), and follow up with the subject regarding any unresolved AEs.

If a subject withdraws consent for the study, no further assessments will be performed. Vertex may retain and continue using the study data and samples after the study ends, and may use the samples and information in the development of the study compound, for other drugs and diagnostics, in publications and presentations, and for education purposes. If a subject withdraws from the study, the study data and samples collected will remain part of the study. A subject will not be able to request the withdrawal of his/her information from the study data. A subject may request destruction of the samples collected from him/her during the study as long as those samples can be identified as his/her samples.

### 9.10 Replacement of Subjects

Subjects who withdraw or are withdrawn during the study drug Treatment Period will not be replaced.

#### 10 STUDY DRUG INFORMATION AND MANAGEMENT

#### 10.1 Preparation and Dispensing

Study drug may be dispensed only under the supervision of the investigator or an authorized designee and only for administration to the study subjects. An interactive web response system (IWRS) will be used to dispense dosage based on subject weight and age.

### 10.2 Packaging and Labeling

Study drug tablets will be supplied in blister cards by Vertex. Study drug labeling will be in compliance with applicable local and national regulations. Additional details regarding packaging, labeling, and dispensing for study drug will be in the Pharmacy Manual.

### 10.3 Study Drug Supply, Storage, and Handling

Table 10-1 provides the study drug information. The investigator, or an authorized designee (e.g., a licensed pharmacist), will ensure that all investigational product is stored in a secured area, under recommended storage conditions, and in accordance with applicable regulatory requirements. To ensure adequate records, all study drugs will be accounted for via the drug accountability forms as instructed by Vertex.

Detailed instructions regarding the storage, handling, and dispensation of the study drug will be provided in the Pharmacy Manual.

| | Tablet Strength | |
|---|---|---|
| Drug Name, Dosing Form, Route | Subjects 6 to <12 years and <30 kg | Subjects 6 to <12 years and ≥30 kg or ≥12 years |
| ELX/TEZ/IVA, FDC tablet, oral | | |
| ELX | 50 mg | 100 mg |
| TEZ | 25 mg | 50 mg |
| IVA | 37.5 mg | 75 mg |
| IVA, tablet, oral | 75 mg | 150 mg |

Table 10-1 Study Drug: Dosing Form/Route/Strength

ELX: elexacaftor; FDC: fixed-dose combination; IVA: ivacaftor; TEZ: tezacaftor

Note: See Table 9-3 for details on study drug administration.

### 10.4 Drug Accountability

The pharmacist or designated study site staff will maintain information about the dates and amounts of (1) study drug received; (2) study drug dispensed to the subjects; and (3) study drug returned by the subjects. Subjects will be instructed to return all used and unused materials associated with the study drug to the site. These materials will be retained at the site according to instructions provided by Vertex or its designee. The study monitor will review study drug records and inventory throughout the study. If a site uses a site-specific drug accountability system and/or process, including processes associated with the destruction of returned materials, the process must be documented and approved by Vertex. The study monitor must review the drug accountability documentation on a regular basis. The study monitor will promptly communicate to Vertex any discrepancies he or she is unable to resolve with the site.

### 10.5 Disposal, Return, or Retention of Unused Drug

The study site staff or pharmacy personnel will retain all materials returned by the subjects until the study monitor has performed drug accountability. The investigator will ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Vertex. Destruction will be adequately documented.

The principal investigator, study site staff, including pharmacy personnel will assist Vertex with any recall activities (as applicable) and place impacted investigational medicinal product (IMP) in quarantine when requested.

### 10.6 Compliance

To ensure treatment compliance, the investigator or designee will supervise all study drug dosing that occurs at the site. At each visit, site personnel will review that the subject is compliant with study drug dosing and remind the subject of study drug dosing requirements. Compliance will also be assessed by ongoing study drug count.

If a subject demonstrates continued noncompliance of study drug dosing despite educational efforts, the investigator should consider discontinuing the subject from the study.

### 10.7 Blinding and Unblinding

This is an open-label study; however, subjects and their legally appointed and authorized representative (e.g., parent or legal guardian) should not be informed of their study-related SwCl,

LCI, and spirometry results until the study has been completed, regardless if the subject permanently discontinues treatment. In addition, the Vertex study team will not have access to the SwCl, LCI, or spirometry of the present study until the data lock of the parent study.

#### 11 ASSESSMENTS

The schedule of assessments is shown in Table 3-1.

The following assessments must be performed in the order specified below when more than 1 assessment is required at a particular time point:

- 1. The CFQ-R should be completed before the start of any other assessments (except signing of ICF or assent) scheduled at that visit.
- 2. The MBW assessment should be performed before spirometry.

### 11.1 Subject and Disease Characteristics

Subject and disease characteristics include the following: demographics, medical history, height, and weight. Select demographic and medical history will be derived from the parent study.

#### 11.2 Efficacy and Pharmacodynamics

#### 11.2.1 Sweat Chloride

The sweat chloride test is a standard diagnostic tool for CF, serving as a biomarker of CFTR activity. Sweat samples will be sent to a central laboratory for testing and interpretation of results. Individual sweat chloride test results will not be disclosed to the study sites. Specific instructions for collection, handling, processing, and shipping of sweat chloride samples to the central laboratory will be provided separately. The sweat chloride test must be conducted predose relative to the morning dose of study drug during the Treatment Period. At each time point, 2 samples will be collected, 1 sample from each arm (left and right).

See Section 10.7 for information about access to SwCl results.

#### 11.2.2 Multiple-breath Washout

The N<sub>2</sub>-MBW testing will be performed in multiple replicates for each visit and the final LCI value will be calculated from the technically acceptable washout replicates by a central reader. The final LCI value at each visit will be the value provided by the LCI vendor based on the replicates.

At all visits, all MBW tests should be performed pre-bronchodilator as described in Section 11.2.3. The MBW should be performed before the spirometry assessment (Section 11). See Section 10.7 for information about access to LCI results.

#### 11.2.3 Spirometry

Spirometry will be performed according to the American Thoracic Society Guidelines/European Respiratory Society Guidelines<sup>12</sup> and according to the additional guidelines that follow.

Pre-bronchodilator spirometry is defined as spirometry testing performed for subjects who have

• withheld their short-acting bronchodilators (e.g., albuterol) or anticholinergic (e.g., ipratropium bromide [Atrovent®]) for more than 4 hours before the spirometry assessment;

- withheld their long-acting bronchodilator (e.g., salmeterol) for more than 12 hours before the spirometry assessment; and
- withheld their once-daily, long-acting bronchodilator (e.g., tiotropium bromide [Spiriva®]) for more than 24 hours before the spirometry assessment.

At all visits, all spirometry assessments should be performed pre-bronchodilator. During the Treatment Period, spirometry assessments must be performed before study drug dosing (Section 9.6.1) at approximately the same time at each visit. In the event that a subject forgets to withhold bronchodilator(s), spirometry should be performed according to the following:

- If a subject's Day 1 spirometry assessment is pre-bronchodilator, but, on a subsequent visit, the subject forgets to withhold bronchodilator use, a post-bronchodilator spirometry assessment will be obtained for that visit only, and the visit will not be rescheduled.
- If, on Day 1, the subject forgets to withhold his/her dose of bronchodilator, spirometry should be performed post-bronchodilator, and all subsequent spirometric measurements (according to the schedule of assessments) should be performed post-bronchodilator.
- Each spirometry assessment will be recorded in the source documents as pre- or post-bronchodilator.

All sites will be provided with spirometers to be used for all study assessments. Spirometry data will be transmitted to a centralized spirometry service for quality review.

See Section 10.7 for information about access to spirometry results.

The measured spirometric values listed below will be converted to percent predicted values using the standard equations of the Global Lung Function Initiative (GLI).<sup>13</sup>

- FEV<sub>1</sub> (L)
- Forced vital capacity (FVC) (L)
- FEV<sub>1</sub>/FVC (ratio)
- Forced expiratory flow, midexpiratory phase (FEF<sub>25%-75%</sub>) (L/s)

### 11.2.4 Cystic Fibrosis Questionnaire-Revised

The questionnaires provide information about demographics; general quality of life, school, work, or daily activities; and symptom difficulties (pertaining to CF).

Subjects/caregivers will be asked to complete the CFQ-R in their native language, if validated translations are available.<sup>14, 15</sup> If there is no validated translation available in the subject's native language, the subject will not complete the questionnaire. Copies of the CFQ-R used will be provided in the Study Reference Manual. Validated translations of the CFQ-R, if available, will be provided for participating centers in non-English-speaking countries.<sup>16, 17</sup>

The CFQ-R will be completed before any other assessments are performed at that visit.

#### 11.3 Other Assessments

#### 11.3.1 Blood Biomarkers

Blood samples for blood biomarker analysis will be collected and banked for potential exploratory evaluation of correlations between blood biomarkers (e.g., proteins, peptides, lipids, vitamins, endogenous metabolites, and RNA) with PD, treatment benefit, and AEs.

Specific instructions for the collection, processing, storage, and shipment of blood biomarker samples will be provided in the Laboratory Manual.

### 11.4 Safety

Safety evaluations will include AEs, clinical laboratory assessments, clinical evaluation of ECGs, vital signs, height, weight, pulse oximetry, physical examinations (PEs), and ophthalmologic examinations.

#### 11.4.1 Adverse Events

All AEs will be assessed, documented, and reported in accordance with current ICH E6 GCP Guidelines. Section 13.1 outlines the definitions, collection periods, criteria, and procedures for documenting, grading, and reporting AEs. Electronic AE case report form (CRF) completion guidelines for investigators as well as training will be provided.

### 11.4.2 Clinical Laboratory Assessments

Blood and urine samples will be analyzed at a central laboratory, with the exception of the urine pregnancy tests. As described below, urine pregnancy tests will either be analyzed by the site or at home using a home kit. On Day 1, blood samples will be collected before the first dose of the study drug. Specific instructions for the collection, processing, and shipment of samples will be provided in a separate Laboratory Manual.

Laboratory test results that are abnormal and considered clinically significant will be reported as AEs (see Section 13.1).

The safety laboratory test panels are shown in Table 11-1.

Table 11-1 Safety Laboratory Test Panels

| Serum Chemistry | Hematology | Urinalysis <sup>a</sup> |
|---|---|---|
| Glucose | Hemoglobin | Leukocyte esterase |
| Blood urea nitrogen <sup>b</sup> | Erythrocytes | Nitrite |
| Creatinine | Mean corpuscular volume | Urobilinogen |
| Sodium | Platelets | Urine protein |
| Potassium | Reticulocytes | pН |
| Calcium | Leukocytes | Urine blood |
| Chloride | Differential (absolute and percent): | Specific gravity |
| Magnesium | Eosinophils | Urine ketones |
| Bicarbonate | Basophils | Urine bilirubin |
| Phosphate | Neutrophils | Urine glucose |
| Total bilirubin, direct bilirubin, | Lymphocytes | |
| indirect bilirubin | Monocytes | |
| Alkaline phosphatase | Coagulation | |
| Aspartate transaminase | Activated partial thromboplastin time | |
| Alanine transaminase | Prothrombin time | |
| Amylase | Prothrombin time International | |
| Lipase | Normalized Ratio | |
| Gamma-glutamyl transferase | | |
| Protein | | |
| Albumin | | |
| Creatine kinase | | |
| Cholesterol | | |

<sup>&</sup>lt;sup>a</sup> If urinalysis results are positive for leukocyte esterase, nitrite, protein, or blood, microscopic examination of urine will be done, and results will be provided for leukocytes, crystals, bacteria, and casts.

Pregnancy ( $\beta$ -human chorionic gonadotropin) Tests for all Female Subjects: All female subjects must have a pregnancy test every 4 weeks. Serum pregnancy tests will be performed at the study site and analyzed at the central laboratory. Urine pregnancy tests will be performed and analyzed at the site or, at assessment time points when telephone contact takes the place of a clinic visit, at home by using a home kit provided by the study site. Results of a home urine pregnancy test will be reported to the site by telephone. The urine pregnancy test on Day 1 must be negative before the first dose of study drug is administered to the subject. Additional pregnancy tests may be required according to local regulations and/or requirements.

Additional Evaluations: Additional clinical laboratory evaluations will be performed at other times if judged by the investigator to be clinically appropriate.

For the purposes of study conduct and unless noted otherwise, only laboratory tests done in the central laboratory may be used. Local laboratories may be used at the discretion of the local investigator for management of urgent medical issues. If a local laboratory test value is found to be abnormal and clinically significant, it will be verified by the central laboratory as soon as possible after the investigator becomes aware of the abnormal result. If it is not possible to send a timely specimen to the central laboratory (e.g., the subject was hospitalized elsewhere), the investigator may base the assessment of an AE on the local laboratory value.

b If blood urea nitrogen cannot be collected, urea may be substituted.

### 11.4.3 Physical Examinations and Vital Signs

A PE of all body systems and vital signs assessment will be performed at select study visits. At other visits, symptom-directed PEs and symptom-directed vital signs assessments can be performed at the discretion of the investigator or healthcare provider.

A PE includes a review of the following systems: head, neck, and thyroid; eyes, ears, nose, and throat (EENT); respiratory; cardiovascular; lymph nodes; abdomen; skin; musculoskeletal; and neurological. Breast, anorectal, and genital examinations will be performed when medically indicated. After screening, any clinically significant abnormal findings in PEs will be reported as AEs.

Vital signs include blood pressure (systolic and diastolic), temperature, pulse rate, and respiration rate. The subject will be instructed to rest for at least 5 minutes before vital signs are assessed.

Arterial oxygen saturation by pulse oximetry will be assessed following at least a 5-minute rest and before study drug dosing.

### 11.4.4 Height and Weight

Height and weight will be measured with shoes off.

### 11.4.5 Electrocardiograms

Standard 12-lead ECGs will be performed using a machine with printout. Additional standard 12-lead ECGs will be performed at any other time if clinically indicated. The performance of all ECGs will adhere to the following guidelines:

- The ECG will be done before any other procedures that may affect heart rate, such as blood draws
- The subject will be instructed to rest for at least 5 minutes before having an ECG

A printout of the ECG traces will be made for safety review by the investigator and maintained with source documentation. Clinically significant ECG abnormalities occurring during the study through the Safety Follow-up Visit will be recorded as AEs.

To ensure safety of the subjects, a qualified individual at the study site will make comparisons to baseline measurements. If the QTcF is increased by >60 msec from the baseline or an absolute QTcF value is ≥500 msec for any scheduled ECG, 2 additional ECGs will be performed approximately 2 to 4 minutes apart to confirm the original measurement. If either of the QTcF values from these repeated ECGs remains above the threshold value (>60 msec from baseline or ≥500 msec), a single ECG will be repeated at least hourly until QTcF values from 2 successive ECGs fall below the threshold value that triggered the repeat measurement.

### 11.4.6 Ophthalmologic Examination

Ophthalmologic examinations do not need to be completed if there is documentation of bilateral lens removal for the subject.

All examinations will be conducted by a licensed ophthalmologist or optometrist and will include:

• measurement of best-corrected distance visual acuity of each eye; and

• pharmacologically dilated examination of the lens with a slit lamp.

Ophthalmologic examinations are required at select study visits in the Treatment Period (Table 3-1). These examinations should be completed within the specified 4-week window around the relevant study visit. A single ophthalmologic examination is required at completion of study participation (defined in Section 9.1.5); this examination should be completed within 4 weeks prior to the last study visit except for subjects who have withdrawn consent or assent. Ophthalmologic examinations are only required if the cumulative study drug exposure (in the parent study and current study) is at least 12 weeks since the last study ophthalmologic examination.

Any clinically significant abnormal findings will be reported as AEs.

### 11.4.7 Contraception and Pregnancy

The effects of ELX monotherapy or in combination with TEZ/IVA on conception, pregnancy, and lactation in humans are not known. ELX, TEZ, and IVA did not show genotoxic potential in a standard battery of in vitro (Ames test, chromosomal aberration, or micronucleus in cultured mammalian cells) and in vivo (rodent micronucleus) studies. Reproductive toxicology studies of ELX, TEZ, and IVA have not shown teratogenicity in rats and rabbits.

### 11.4.7.1 Contraception

#### Contraception requirement is waived for the following:

- True abstinence for the subject, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception. True abstinence must be practiced from the date of informed consent through 90 days after the last dose of study drug.
- If the subjects is male and is infertile (e.g., bilateral orchiectomy). If a male subject is assumed to have complete bilateral absence of the vas deferens, infertility must be documented before the first dose of study drug (e.g., examination of a semen specimen or by demonstration of the absence of the vas deferens by ultrasound).
- If the subject is female is of non-childbearing potential. To be considered of non-childbearing potential, the female must meet at least 1 of the following criteria:
  - o Postmenopausal: Amenorrheic for at least 12 consecutive months and a serum follicle-stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females
  - o Documented hysterectomy or bilateral oophorectomy/salpingo-oophorectomy
  - o Note: All other females (including females with tubal ligations) will be considered to be of childbearing potential.
- Same-sex relationships

For subjects for whom the contraception requirement is not waived, study participation requires a commitment from the subject that <u>at least 1 acceptable method</u> of contraception is used. Methods of contraception must be in successful use from signing of consent (or assent, when applicable), approximately 28 days before the first dose of study drug (unless otherwise

noted), and until 90 days following the last dose of study drug. Additional contraception requirements may need to be followed according to local regulations and/or requirements. Acceptable methods of contraception are listed in Table 11-2.

**Table 11-2** Acceptable Methods of Contraception

| | Male Subjects and<br>Their Female<br>(Non-study) Partners | Female Subjects and<br>Their Male (Non-study)<br>Partners |
|---|---|---|
| Vasectomy performed at least 6 months previously, with a documented negative postvasectomy semen analysis for sperm | Yes | Yes |
| Bilateral tubal occlusion (e.g., ligation) performed at least 6 months previously | Yes | Yes |
| Male or female condom with or without spermicide <sup>a</sup> | Yes | Yes |
| Female barrier contraception (such as diaphragm, cervical cap, or sponge) with spermicide | Yes | Yes |
| Continuous use of an intrauterine device for at least 90 days before the first dose of study drug | | |
| Hormone-releasing | Yes | Yes |
| Non-hormone releasing | Yes | Yes |
| Oral, implanted, injected, or vaginal <b>hormonal</b> contraceptives, if successfully used for at least 60 days before the first dose of study drug | Yes | Yes |

<sup>&</sup>lt;sup>a</sup> A female condom cannot be used with a male condom due to risk of tearing.

#### Additional notes:

- If over the course of the study the subject meets the criteria for waiving the contraception requirements, the subject does not need to follow the contraceptive methods listed in Table 11-2.
- If over the course of the study the subject's status changes and the subject does not meet the criteria for waiving the contraception requirements, the subject must begin following the contraceptive methods listed in Table 11-2.
- Male subjects must not donate sperm during the period starting from the first dose of study drug until 90 days after the last dose of study drug.
- Female subjects should not nurse a child during the period starting from the first dose of study drug until 90 days after the last dose of study drug.
- Female partners of male subjects should not plan to become pregnant during the study or within 90 days after the last dose of study drug, with the exception of those who plan to become pregnant by artificial insemination using sperm banked by the male subject before the first dose of study drug or sperm from another source.

### 11.4.7.2 **Pregnancy**

Subjects will be counseled to inform the investigator of any pregnancy that occurs during study treatment and for 90 days after the last dose of study drug.

If a subject, or the female partner of a male subject, becomes pregnant while participating in the study, the study drug will be permanently discontinued immediately. The investigator will 1) notify the medical monitor and Vertex Global Patient Safety (GPS) within 24 hours of the site's knowledge of the subject's (or partner's) pregnancy, and 2) send the Pregnancy Information Collection Form to Vertex GPS. Male subjects with female partners who become pregnant during the study must use a male condom to avoid exposure of a potential embryo or fetus to study drug via the seminal fluid.

The subject or partner will be followed until the end of the pregnancy and the infant will be followed for 1 year after the birth, provided informed consent (and assent, as applicable) is obtained. A separate ICF will be provided to explain these follow-up activities. Pregnancy itself does not constitute an AE.

#### 12 STATISTICAL ANALYSIS

This section presents a summary of the planned analyses for this protocol. Statistical analysis details will be provided in the statistical analysis plan (SAP), which will be finalized before the clinical data lock for the study.

### 12.1 Sample Size

The primary objective of the study is the evaluation of the long-term safety and tolerability of ELX/TEZ/IVA. This is an open-label extension study that will enroll subjects who did not discontinue study drug during the Treatment Period in the parent study and meet eligibility criteria in this study.

Approximately 108 subjects are expected to enroll in this extension study.

# 12.2 Analysis Sets

The **Open-label All Subjects Set** is defined as all subjects who were enrolled (defined as subject having data in the clinical database) in this open-label study. This analysis set will be used for individual subject data listings and disposition summary tables unless otherwise specified.

The **Open-label Full Analysis Set (OL-FAS)** is defined as all enrolled subjects who have received at least 1 dose of study drug in this open-label study. The OL-FAS will be used to summarize subject demographics and baseline characteristics and for all efficacy analyses unless otherwise specified.

The **Open-label Safety Set (OL-SS)** is defined as all subjects who have received at least 1 dose of study drug in this open-label study. The OL-SS will be used for all safety analyses unless otherwise specified.

### 12.3 Statistical Analysis

This section presents a summary of the planned analyses for this protocol. Statistical analysis details will be provided in the statistical analysis plan (SAP), which will be finalized before the clinical data lock for the study.

#### 12.3.1 General Considerations

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, SD, median, minimum value (min), and maximum value (max).

Categorical variables will be summarized using counts and percentages.

The **baseline value**, unless otherwise specified, for the long-term safety analysis will be the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of ELX/TEZ/IVA either in the parent study or the open label study, as applicable. The baseline value for the long-term efficacy analysis will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the parent study. For assessments collected in duplicate or triplicate, the baseline will be defined as the average of non-missing values.

Change (absolute change) from baseline will be calculated as <u>Post-baseline value – Baseline</u> value.

The **Efficacy Analysis Period** in the open-label study will include the time from the first dose of study drug in the open-label study to the last scheduled efficacy visit in the open-label study, unless otherwise specified.

The **Treatment-emergent (TE) Period** in the open-label study will include the time from the first dose of study drug in the open-label study to 28 days after the last dose of the study drug in the open-label study or to the completion date of study participation (as defined in Section 9.1.5), whichever occurs first.

#### 12.3.2 Background Characteristics

### 12.3.2.1 Subject Disposition

Subject disposition will be summarized for the Open-label All Subjects Set. The number and percentage of subjects in the following categories will be summarized as appropriate:

- Open-label All Subjects Set
- Dosed (OL-SS)
- Enrolled and dosed (OL-FAS)
- Completed Treatment Period
- Prematurely discontinued treatment and the reasons for discontinuation
- Completed study
- Prematurely discontinued the study and the reasons for discontinuation

#### 12.3.2.2 Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized by descriptive summary statistics. Demographics and baseline characteristics will be obtained from the parent study baseline.

The following demographics and baseline characteristics will be summarized for the OL-SS and will include (but are not limited to) sex, race, age, baseline weight, baseline height, and baseline body mass index (BMI).

Medical history will be summarized by MedDRA System Organ Class (SOC) and Preferred Term (PT) for the OL-SS.
# 12.3.2.3 Prior and Concomitant Medications

Medications used will be coded using the World Health Organization-Drug Dictionary and categorized as the following:

- **Prior medication:** any medication that was administered within the 56 days before the first dose of study drug in this open-label study
- **Concomitant medication:** medication continued or newly received during the TE Period in this open-label study
- **Post-treatment medication:** medication continued or newly received after the TE Period in this open-label study

A given medication may be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment. If a medication has a missing or partially missing start/end date or time and if it cannot be determined whether it was taken before initial dosing, concomitantly during the TE Period, or beyond the TE Period, it will be considered in all 3 categories of prior, concomitant, and post-treatment medication.

Prior medications and concomitant medications will be summarized descriptively by Preferred Name based on the OL-SS. Post-treatment medications will be provided separately in an individual subject data listing.

# 12.3.2.4 Study Drug Exposure and Compliance

Study drug exposure will be summarized based on the OL-SS, defined as the last day of study drug in this open-label study minus the first day of study drug in this open-label study plus 1, regardless of study drug interruption.

Study drug compliance will be summarized based on the OL-FAS and will be calculated as:  $100 \times [1 - (\text{total number of days of study drug interruption in this open-label study}) / (duration of study drug exposure in days in this open-label study)]. A study drug interruption on a given day is defined as an interruption of any study drug on that day.$ 

In addition, percentage of tablets taken in the open-label study will also be summarized based on the OL-FAS, and will be calculated as  $100 \times [(\text{total number of tablets dispensed in the open-label study}) - ((\text{total number of tablets returned in the open-label study})] / ((total number of tablets planned to be taken per day × duration of study drug exposure in days for the open-label study).$ 

# 12.3.2.5 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being.

All IPDs will be provided in an individual subject data listing, as appropriate.

# 12.3.3 Efficacy Analysis

The secondary objectives of the study are the evaluation of the efficacy and PD of ELX/TEZ/IVA.

# 12.3.3.1 Analysis of Primary Efficacy and Pharmacodynamic Endpoints

Not applicable, as efficacy and PD are not primary objectives.

#### 12.3.3.2 Analysis of Secondary Efficacy and Pharmacodynamic Endpoints

The Secondary Endpoints include:

#### • Absolute change from baseline in SwCl

The analysis of this endpoint will be performed using a mixed-effects model for repeated measures (MMRM) with absolute change from baseline in SwCl at each post-baseline visit in this current open-label study as the dependent variable. The model will include the parent study treatment group, visit, and parent study treatment-by-visit interaction as fixed effects, and will be adjusted for main covariates as appropriate. The least squares (LS) mean estimate with a 2-sided 95% CI at each visit will be provided.

#### • Absolute change from baseline in LCI<sub>2.5</sub>

Analysis of this efficacy endpoint will be based on a MMRM model similar to the analysis of the absolute change from baseline in SwCl.

# 12.3.3.3 Analysis of Other Efficacy and Pharmacodynamic Endpoints

Other Endpoints include:

#### • Absolute change from baseline in ppFEV<sub>1</sub>

Analysis of this variable will be based on an MMRM model similar to the analysis of the absolute change from baseline in LCI<sub>2.5</sub>.

# • Absolute change from baseline in CFQ-R respiratory domain score

Analysis of this variable will be based on an MMRM model similar to the analysis of the absolute change from baseline in LCI<sub>2.5</sub>.

#### 12.3.3.4 Multiplicity Adjustment

No multiplicity adjustment is planned.

#### 12.3.4 Safety Analysis

The primary objective of the study is the evaluation of the long-term safety and tolerability of ELX/TEZ/IVA. All safety analyses will be based on the TE Period in this open-label study for subjects in the OL-SS, unless otherwise specified.

The overall safety profile of study drug will be assessed in terms of the following safety and tolerability endpoints:

- Incidence of treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (i.e., serum chemistry, hematology, coagulation, and urinalysis)
- ECGs
- Vital signs
- Pulse oximetry

In general, long term safety analysis will be performed in a pooled fashion. All safety data will be presented in individual subject data listings. Only descriptive analyses of safety data will be performed.

# 12.3.4.1 Adverse Events

For analysis purposes, AEs will be classified as pretreatment AEs, TEAEs, or post-treatment AEs, defined as follows:

- **Pretreatment AE**: any AE that occurred since the end of the TE Period in the parent study and before the first dose of ELX/TEZ/IVA in the TE Period in the open-label study
- **TEAE**: any AE that worsened (either in severity or seriousness) or newly developed at or after the first dose date of ELX/TEZ/IVA in the TE Period in this open-label study
- **Post-treatment AE**: any AE that worsened (either in severity or seriousness) or newly developed after the TE Period in this open-label study

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after study drug treatment, then the AEs will be classified as TEAEs.

AE summary tables will be presented for TEAEs only and will include the following:

- All TEAEs
- TEAEs by strongest relationship
- TEAEs by maximum severity
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- Serious TEAEs
- TEAEs leading to death
- Grade 3 and Grade 4 TEAEs
- Frequently reported TEAEs

Summaries will be presented by MedDRA SOC and PT using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries.

Listings containing individual subject level AE data will be provided separately for:

- Serious TEAEs
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- TEAEs leading to death

In addition, all AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings

# 12.3.4.2 Clinical Laboratory Assessments

For the TE laboratory measurements, the observed values and change from baseline values of the continuous laboratory parameters will be summarized in SI units at each time point during the TE Period.

For threshold analysis, the number and percentage of subjects with at least 1 threshold event during the TE Period will be summarized. The threshold criteria and selected parameters will be provided in the SAP.

Results of urinalysis and pregnancy tests will be listed in individual subject data listings only. In addition, a listing containing individual subject laboratory assessment values will be provided. This listing will include data from scheduled and unscheduled time points.

Additional safety laboratory data analyses may be described in the SAP.

#### 12.3.4.3 Electrocardiogram

For the TE ECG measurements, a summary of observed values and change from baseline values will be provided at each time point during the TE Period, for the following ECG interval measurements (in msec): RR, PR, QT, QT corrected for heart rate (HR) intervals (QTcF), QRS duration, and HR (beats per minute).

For threshold analysis, the number and percentage of subjects with at least 1 threshold event during the TE Period will be summarized. The threshold criteria will be provided in the SAP.

Additional ECG analyses may be described in the SAP.

# **12.3.4.4** Vital Signs

For the TE vital signs measurements, the observed values and change from baseline values will be summarized at each time point during the TE Period in this open-label study. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

For threshold analysis, the number and percentage of subjects with at least 1 threshold event during the TE Period will be summarized. The threshold criteria will be provided in the SAP.

Additional vital signs analyses may be described in the SAP.

#### 12.3.4.5 Pulse Oximetry

For the TE pulse oximetry measurements, a summary of observed values and change from baseline values will be provided at each time point during the TE Period, for the percent of oxygen saturation by pulse oximetry.

# **12.3.4.6** Physical Examination

No tables/figures/listings will be provided for PE data.

#### 12.3.4.7 Other Safety Analyses

Details of other safety analyses may be included in the SAP.

# 12.4 Interim Analysis

Interim analyses may take place at any time at the discretion of the sponsor.

#### 12.5 Data Monitoring Committee Analysis

A data monitoring committee (DMC) will conduct periodic safety review(s) of study data as outlined in the DMC charter.

# 13 PROCEDURAL, ETHICAL, REGULATORY, AND ADMINISTRATIVE CONSIDERATIONS

# 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting

#### 13.1.1 Adverse Events

#### 13.1.1.1 Definition of an Adverse Event

An AE is defined as any untoward medical occurrence in a subject during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or worsening of a pre-existing condition (e.g., increase in its severity or frequency) after the ICF is signed.

An AE is considered serious if it meets the definition in Section 13.1.2.1.

# 13.1.1.2 Clinically Significant Assessments

Study assessments including laboratory tests, ECGs, PEs, and vital signs will be assessed and those deemed to have clinically significant worsening from baseline will be documented as an AE. When possible, a clinical diagnosis for the study assessment will be provided, rather than the abnormal test result alone (e.g., urinary tract infection, anemia). In the absence of a diagnosis, the abnormal study assessment itself will be listed as the AE (e.g., bacteria in urine or decreased hemoglobin).

An abnormal study assessment is considered clinically significant if the subject has 1 or more of the following:

- Concomitant signs or symptoms related to the abnormal study assessment
- Further diagnostic testing or medical/surgical intervention
- A change in the dose of study drug or discontinuation from the study

Repeat testing to determine whether the result is abnormal, in the absence of any of the above criteria, does not necessarily meet clinically significant criteria. The determination of whether the study assessment results are clinically significant will be made by the investigator.

A laboratory value that is Grade 4 will not automatically be an SAE. A Grade 4 laboratory value will be an SAE if the subject's clinical status indicates a life-threatening AE.

#### 13.1.1.3 Documentation of Adverse Events

All AEs will be collected from the time the ICF is signed until the following times:

• For subjects who do not enroll: until time of screen failure (e.g., screen failure, withdrawal of consent)

- For enrolled subjects who have a Safety Follow-up Visit: through the Safety Follow-up Visit
- For enrolled subjects who do not have a Safety Follow-up Visit, the earliest of
  - o 28 days after the last dose of study drug, or
  - o the ETT Visit, if that visit is 3 weeks or later following the last dose of study drug (see Section 9.1.3)

All subjects' parents or legal guardians will be queried, using nonleading questions, about the occurrence of AEs at each study visit. When possible, a constellation of signs and/or symptoms will be identified as 1 overall event or diagnosis. All AEs for enrolled subjects will be recorded in the CRF and source document. AEs for subjects who are screened but not subsequently enrolled will be recorded only in the subject's source documents. The following data will be documented for each AE:

- Description of the event
- Classification of "serious" or "nonserious"
- Date of first occurrence and date of resolution (if applicable)
- Severity
- Causal relationship to study drug(s)
- Action taken
- Outcome
- Concomitant medication or other treatment given

# 13.1.1.4 Adverse Event Severity

The investigator will determine and record the severity of all serious and nonserious AEs. The guidance available at the following website will be consulted: Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, Cancer Therapy Evaluation Program, <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm</a> (Accessed September 2019). When considering the severity of an AE in a pediatric subject, the investigator will consider that reference ranges for pediatric clinical laboratory parameters may differ from those in the CTCAE. The severity of an AE described by a term that does not appear in the CTCAE will be determined according to the definitions in Table 13-1.

**Table 13-1** Grading of AE Severity

| Classification | Description |
|---|---|
| Grade 1 (Mild) | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| Grade 2 (Moderate) | Moderate; minimal, local, or noninvasive intervention indicated; limiting age-<br>appropriate instrumental ADL <sup>a</sup> |
| Grade 3 (Severe) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL <sup>b</sup> |
| Grade 4 (Life-threatening) | Life-threatening consequences; urgent intervention indicated |
| Grade 5 (Death) | Death related to adverse event |

Table 13-1 Grading of AE Severity

| Classification | Description | |
|---|---|---|
| Source: http://ctep.canc | .gov/protocolDevelopment/electronic_applications/ctc.htm (Accessed September 2019 | 9) |
| ADL: activities of daily | iving; AE: adverse event | |

Note: A semi-colon indicates 'or' within the description of the grade.

- Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- b Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

# 13.1.1.5 Adverse Event Causality

Every effort will be made by the investigator to assess the relationship of the AE, if any, to the study drug(s). Causality will be classified using the categories in Table 13-2.

**Table 13-2** Classifications for AE Causality

| Classification | Definition |
|---|---|
| Related | There is an association between the event and the administration of investigational study drug, a plausible mechanism for the event to be related to the investigational study drug and causes other than the investigational study drug have been ruled out and/or the event reappeared on re-exposure to the investigational study drug. |
| Possibly related | There is an association between the event and the administration of the investigational study drug and there is a plausible mechanism for the event to be related to investigational study drug, but there may also be alternative etiology, such as characteristics of the subject's clinical status or underlying disease. |
| Unlikely related | The event is unlikely to be related to the investigational study drug and likely to be related to factors other than investigational study drug. |
| Not related | The event is related to an etiology other than the investigational study drug (the alternative etiology will be documented in the subject's medical record). |

AE: adverse event

# 13.1.1.6 Study Drug Action Taken

The investigator will classify the study drug action taken with regard to the AE. The action taken will be classified according to the categories in Table 13-3.

Table 13-3 Classifications for Study Drug Action Taken With Regard to an AE

| Classificationa | Definition |
|---|---|
| Dose not changed | Study drug dose not changed in response to an AE |
| Dose reduced | Study drug dose reduced in response to an AE |
| Drug interrupted | Study drug administration interrupted in response to an AE |
| Drug withdrawn | Study drug administration permanently discontinued in response to an AE |
| Not applicable Action taken regarding study drug administration does not apply. | |
| | "Not applicable" will be used in circumstances such as when the investigational |
| | treatment had been completed before the AE began and no opportunity to decide |
| | whether to continue, interrupt, or withdraw treatment is possible. |

AE: adverse event

<sup>&</sup>lt;sup>a</sup> Refer to Sections 9.6.1 and 9.8 for directions regarding what drug actions are permitted per protocol.

#### 13.1.1.7 Adverse Event Outcome

An AE will be followed until the investigator has determined and provided the final outcome. The outcome will be classified according to the categories in Table 13-4.

Table 13-4 Classifications for Outcome of an AE

| Classification | Definition |
|---|---|
| Recovered/resolved | Resolution of an AE with no residual signs or symptoms |
| Recovered/resolved with sequelae | Resolution of an AE with residual signs or symptoms |
| Not recovered/not resolved (continuing) | Either incomplete improvement or no improvement of an AE, such that it remains ongoing |
| Fatal | Outcome of an AE is death. "Fatal" will be used when death is at least possibly related to the AE. |
| Unknown | Outcome of an AE is not known (e.g., a subject lost to followup) |

AE: adverse event

#### 13.1.1.8 Treatment Given

The investigator ensures adequate medical care is provided to subjects for any AEs, including clinically significant laboratory values related to study drug. In addition, the investigator will describe whether any treatment was given for the AE. "Yes" is used if any treatment was given in response to an AE, and may include treatments such as other medications, surgery, or physical therapy. "No" indicates the absence of any kind of treatment for an AE.

#### 13.1.2 Serious Adverse Events

#### 13.1.2.1 Definition of a Serious Adverse Event

An SAE is any AE that meets any of the following outcomes:

- Fatal (death, regardless of cause, that occurs during participation in the study or occurs after participation and is suspected of being a delayed toxicity due to administration of the study drug)
- Life-threatening, such that the subject was at immediate risk of death from the reaction as it occurred
- Inpatient hospitalization or prolongation of hospitalization
- Persistent or significant disability/incapacity (disability is defined as a substantial disruption of a person's ability to conduct normal life functions)
- Congenital anomaly or birth defect
- Important medical event that, based upon appropriate medical judgment, may jeopardize the subject or may require medical or surgical intervention to prevent 1 of the outcomes listed above (e.g., an allergic bronchospasm requiring intensive treatment in an emergency room or at home)

If a subject has a hospitalization or procedure (e.g., surgery) for an event or condition that occurred before the subject signed the ICF, and the hospitalization or procedure was planned before the subject signed the ICF, the hospitalization or procedure will not be considered to

indicate an SAE, unless an AE caused the hospitalization or procedure to be rescheduled sooner or to be prolonged relative to what was planned. In addition, hospitalizations clearly not associated with an AE (e.g., social hospitalization for purposes of respite care) will not be considered to indicate an SAE.

Clarification will be made between the terms "serious" and "severe" because they are not synonymous. The term "severe" is often used to describe the intensity (severity) of a specific event, as in mild, moderate, or severe myocardial infarction. The event itself, however, may be of relatively minor medical significance, such as a severe headache. This is not the same as "serious", which is based on subject/event outcome or action described above, and is usually associated with events that pose a threat to a subject's life or functioning. Seriousness, not severity, serves as a guide for defining expedited regulatory reporting obligations.

# 13.1.2.2 Reporting and Documentation of Serious Adverse Events

All SAEs that occur after obtaining informed consent through the Safety Follow-up Visit, regardless of causality, will be reported by the investigator to Vertex GPS within 24 hours of identification. In addition, all SAEs that occur after the Safety Follow-up Visit and are considered related to study drug(s) will be reported to Vertex GPS within 24 hours of identification.

For SAEs that occur after obtaining informed consent through the Safety Follow-up Visit, the SAE Form will be completed for new/initial events as well as to report follow-up information on previously reported events. Investigators are asked to report follow-up information as soon as it becomes available to ensure timely reporting to health authorities.

Please send completed SAE Forms to Vertex GPS via:

Email: globalpatientsafety@vrtx.com (preferred choice)

Fax: +1-617-341-6159

For technical issues related to submitting the form, contact telephone: +1-617-341-6677

SAEs that occur after the Safety Follow-up Visit and are considered related to study drug(s) will be recorded on the Vertex Clinical Trial Safety Information Collection Form (hereafter referred to as the "SAE Form") using a recognized medical term or diagnosis that accurately reflects the event. SAEs will be assessed by the investigator for relationship to the investigational study drug(s) and possible etiologies. On the SAE Form, relationship to study drug(s) will be assessed only as related (includes possibly related) or not related (includes unlikely related), and severity assessment will not be required. For the purposes of study analysis, if the event has not resolved at the end of the study reporting period, it will be documented as ongoing. For purposes of regulatory safety monitoring, the investigator is required to follow the event to resolution and report the outcome to Vertex using the SAE Form.

#### 13.1.2.3 Expedited Reporting and Investigator Safety Letters

Vertex, as study sponsor, is responsible for reporting suspected, unexpected, serious adverse reactions (SUSARs) involving the study drug(s) to all regulatory authorities, IEC, and participating investigators in accordance with current ICH E2A Guidelines and/or local regulatory requirements, as applicable. In addition, Vertex, or authorized designee, will be responsible for the submission of safety letters to central IECs.

It is the responsibility of the investigator or designee to promptly notify the local IRB/ IEC of all unexpected serious adverse drug reactions involving risk to human subjects.

# 13.2 Administrative Requirements

# 13.2.1 Product Complaints

A product complaint is defined as any verbal or written communication addressed to Vertex, or designee, of inquiry or dissatisfaction with the identity, strength, quality, or purity of a released drug product, IMP, or medical device. In addition, suspected counterfeit/falsified product is considered a product complaint.

Product complaints are to be reported to Vertex.

#### 13.2.2 Ethical Considerations

The study will be conducted in accordance with the current ICH E6 GCP Guidelines, which are consistent with the ethical principles founded in the Declaration of Helsinki, and in accordance with local applicable laws and regulations. The IRB/IEC will review all appropriate study documentation to safeguard the rights, safety, and well-being of the subjects. The study will be conducted only at sites where IRB/IEC approval has been obtained. The protocol, Investigator's Brochure, sample ICF, advertisements (if applicable), written information given to the subjects (including diary cards), safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB/IEC by the investigator or Vertex, as allowable by local applicable laws and regulations.

# 13.2.3 Subject Information and Informed Consent

After the study has been fully explained, written informed consent will be obtained from the subject or legal representative or guardian (if applicable), and assent will be obtained from the subject (if applicable), before study participation. The method of obtaining and documenting the informed consent and assent (if applicable) and the contents of the consent will comply with current ICH E6 GCP Guidelines and all applicable laws and regulations and will be subject to approval by Vertex or its designee.

#### 13.2.4 Investigator Compliance

No modifications to the protocol will be made without the approval of both the investigator and Vertex. Changes that significantly affect the safety of the subjects, the scope of the investigation, or the scientific quality of the study will require IRB/IEC notification before implementation, except where the modification is necessary to eliminate an apparent immediate hazard to human subjects. Vertex will submit all protocol modifications to the required regulatory authorities.

When circumstances require an immediate departure from procedures set forth in the protocol, the investigator will contact Vertex to discuss the planned course of action. If possible, contact will be made before the implementation of any changes. Any departures from the protocol will be fully documented in the source documentation and in a protocol deviation log.

#### 13.2.5 Access to Records

The investigator will make the office and/or hospital records of subjects enrolled in this study available for inspection by Vertex or its representative at the time of each monitoring visit and for audits. The records will also be available for direct inspection, verification, and copying, as required by applicable laws and regulations, by officials of the regulatory health authorities

(FDA and others). The investigator will comply with applicable privacy and security laws for use and disclosure of information related to the research set forth in this protocol.

# 13.2.6 Subject Privacy

To maintain subject confidentiality and to comply with applicable data protection and privacy laws and regulations, all CRFs, study reports, and communications relating to the study will identify subjects by assigned subject numbers, and access to subject names linked to such numbers will be limited to the site and the study physician and will not be disclosed to Vertex. As required by applicable laws and regulations in the countries in which the study is being conducted, the investigator will allow Vertex and/or its representatives access to all pertinent medical records to allow for the verification of data gathered in the CRFs/SAE Forms and the review of the data collection process. The FDA and regulatory authorities in other jurisdictions, including the IRB/IEC, may also request access to all study records, including source documentation, for inspection.

For sites participating in the US, and in accordance with the Health Insurance Portability and Accountability Act (HIPAA) and associated regulations, an executed HIPAA authorization will be obtained by the site from each subject (or the legal representative of the subject) before research activities may begin. Each HIPAA authorization will comply with all HIPAA requirements including authorization allowing the site access to and use of the subject's personally identifiable health information, authorization for the site to disclose such information to Vertex, the FDA, and other parties requiring access under the protocol, and statements as to the purpose for which such information may be used and for how long.

#### 13.2.7 Record Retention

The investigator will maintain all study records according to current ICH E6 GCP Guidelines and/or applicable local regulatory requirement(s), whichever is longest, as described in the Clinical Trial Agreement. If the investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility and Vertex will be notified.

# 13.2.8 Study Termination

At any time, Vertex may terminate this study in its entirety or may terminate this study at any particular site. In addition, for reasonable cause, either the investigators or their IRBs/IECs may terminate the study at their center.

Conditions that may lead to reasonable cause and warrant termination include, but are not limited to:

- Subject or investigator noncompliance
- Unsatisfactory subject enrollment
- Lack of adherence to protocol procedures
- Lack of evaluable and/or complete data
- Potentially unacceptable risk to study subjects
- Decision to modify drug development plan
- Decision by the FDA or other regulatory authority

Written notification that includes the reason for the clinical study termination is required.

### 13.2.9 End of Study

The end of study is defined as the last scheduled visit (or scheduled contact) of the last subject.

# 13.3 Data Quality Assurance

Vertex or its designated representative will conduct a study site visit to verify the qualifications of each investigator, inspect clinical study site facilities, and inform the investigator of responsibilities and procedures for ensuring adequate and correct study documentation per current ICH E6 GCP Guidelines.

The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each subject. Study data for each enrolled subject will be entered into a CRF by study site personnel using a secure, validated, web-based electronic data capture (EDC) application. Vertex will have read-only access to site-entered clinical data in the EDC application.

Instances of missing, discrepant, or uninterpretable data will be queried with the investigator for resolution. Any changes to study data will be made to the CRF and documented in an audit trail, which will be maintained within the clinical database.

#### 13.4 Monitoring

Monitoring and auditing procedures developed or approved by Vertex will be followed to comply with GCP Guidelines. On-site checking of the CRFs/SAE Forms for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed.

The study will be monitored by Vertex or its designee. Monitoring will be done by a representative of Vertex or designee (study site monitor), who will review the CRFs/SAE Forms and source documents per current ICH E6 GCP Guidelines. The study site monitor will ensure that the investigation is conducted according to the protocol design and regulatory requirements.

# 13.5 Electronic Data Capture

Vertex will provide the study sites with secure access to and training on the EDC application sufficient to permit study site personnel to enter or correct information in the CRFs on the subjects for which they are responsible.

A CRF will be completed for each enrolled study subject. It is the investigator's responsibility to ensure the accuracy, completeness, clarity, and timeliness of the data reported in the subject's CRF. Source documentation supporting the CRF data will indicate the subject's participation in the study and will document the dates and details of study procedures, AEs, other observations, and subject status.

The investigator, or designated representative, will complete the CRF as soon as possible after information is collected.

The audit trail entry will show the user's identification information and the date and time of any correction. The investigator will provide formal approval of all the information in the CRFs, including any changes made to them, to endorse the final submitted data for the subjects for whom the investigator is responsible.

Vertex will retain the CRF data and corresponding audit trails. A copy of the final archival CRF in the form of a compact disc (CD) or other electronic media will be placed in the investigator's study file.

# 13.6 Confidentiality and Disclosure

Any and all scientific, commercial, and technical information disclosed by Vertex in this protocol or elsewhere will be considered the confidential and proprietary property of Vertex. The investigator shall hold such information in confidence and shall not disclose the information to any third party except to such of the investigator's employees and staff as have been made aware that the information is confidential and who are bound to treat it as such and to whom disclosure is necessary to evaluate that information. The investigator shall not use such information for any purpose other than determining mutual interest in performing the study and, if the parties decide to proceed with the study, for the purpose of conducting the study.

The investigator understands that the information developed from this clinical study will be used by Vertex in connection with the development of the study drug and other drugs and diagnostics, and therefore may be disclosed as required to other clinical investigators, business partners and associates, the FDA, and other government agencies. The investigator also understands that, to allow for the use of the information derived from the clinical study, the investigator has the obligation to provide Vertex with complete test results and all data developed in the study.

#### 13.7 Publications and Clinical Study Report

### 13.7.1 Publication of Study Results

Vertex is committed to reporting the design and results of all clinical studies in a complete, accurate, balanced, transparent, and timely manner, consistent with Good Publication Practices (GPP3).<sup>18</sup>

**Publication Planning**: Vertex staff along with the lead principal investigators (PIs), the steering committee (SC), and/or the publication committee (PC) will work together to develop a publication plan.

**Authorship**: Authorship of publications will be determined based on the Recommendations for Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals, which states that authorship should be based on the following 4 criteria<sup>19</sup>:

- 1. Substantial contributions to conception and design, acquisition of data, or analysis and interpretation of data;
- 2. Drafting of the article or revising it critically for important intellectual content;
- 3. Final approval of the version to be published; and
- 4. Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

All authors must meet conditions 1, 2, 3, and 4. All persons designated as authors should qualify for authorship, and all those who qualify should be listed. Contributions such as medical writing, enrollment of subjects, acquisition of funding, collection of data, or general supervision of the research group, alone, do not justify authorship.

**Contributors**: Contributors who meet fewer than all 4 of International Committee of Medical Journal Editors (ICMJE) criteria for authorship will not be listed as authors, but their contribution will be acknowledged and specified either as a group (e.g., "study investigators") or individually (e.g., "served as scientific advisor").

**Publication Review**: As required by a separate clinical study agreement, Vertex must have the opportunity to review all publications, including any manuscripts, abstracts, oral/slide presentations, and book chapters regarding this study before submission to congresses or journals for consideration.

# 13.7.2 Clinical Study Report

A clinical study report (CSR), written in accordance with the current ICH E3 Guideline, will be submitted in accordance with local regulations.

#### 14 REFERENCES

- 1 Cystic Fibrosis Foundation. What is cystic fibrosis? Available at: https://www.cff.org/What-is-CF/About-Cystic-Fibrosis/. Accessed 22 March 2018.
- 2 Cystic Fibrosis Foundation. 2018 Patient Registry Annual Data Report. Bethesda, MD: 2019.
- 3 European Cystic Fibrosis Society. 2017 ECFS Patient Registry Annual Data Report. Karup, Denmark: 2019.
- 4 Rommens JM, Iannuzzi MC, Kerem B, Drumm ML, Melmer G, Dean M, et al. Identification of the cystic fibrosis gene: chromosome walking and jumping. Science. 1989;245(4922):1059-65.
- 5 Kreindler JL. Cystic fibrosis: exploiting its genetic basis in the hunt for new therapies. Pharmacol Ther. 2010;125(2):219-29.
- Konstan MW, McKone EF, Moss RB, Marigowda G, Tian S, Waltz D, et al. Assessment of safety and efficacy of long-term treatment with combination lumacaftor and ivacaftor therapy in patients with cystic fibrosis homozygous for the F508del-CFTR mutation (PROGRESS): a phase 3, extension study. Lancet Respir Med. 2017;5(2):107-18.
- Sawicki GS, McKone E, Pasta DJ, Wagener J, Johnson C, Konstan MW. The effect of ivacaftor on the rate of lung function decline in CF patients with a G551D-CFTR mutation. J Cyst Fibros. 2014;13:S6.
- 8 Horsley A. Lung clearance index in the assessment of airways disease. Respir Med. 2009;103(6):793-99.
- 9 Sinhal S, Galati J, Baldwin DN, Stocks J, Pillow JJ. Reproducibility of multiple breath washout indices in the unsedated preterm neonate. Pediatr Pulmonol. 2010;45(1):62-70.
- Lum S, Gustafsson P, Ljungberg H, Hulskamp G, Bush A, Carr SB, et al. Early detection of cystic fibrosis lung disease: multiple-breath washout versus raised volume tests. Thorax. 2007;62(4):341-47.
- Gustafsson PM, De Jong PA, Tiddens HA, Lindblad A. Multiple-breath inert gas washout and spirometry versus structural lung disease in cystic fibrosis. Thorax. 2008;63(2):129-34.
- Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J. 2005;26(2):319-38.
- Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3–95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.
- Goss CH, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac Soc. 2007;4(4):378-86.
- Ouittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of the Cystic Fibrosis Questionnaire in the United States. Chest. 2005;128(4):2347-54.
- Henry B, Aussage P, Grosskopf C, Goehrs JM. Development of the Cystic Fibrosis Questionnaire (CFQ) for assessing quality of life in pediatric and adult patients. Qual Life Res. 2003;12(1):63-76.
- Wenninger K, Aussage P, Wahn U, Staab D, German Cystic Fibrosis Questionnaire study group. The revised German Cystic Fibrosis Questionnaire: validation of a disease-specific health-related quality of life instrument. Qual Life Res. 2003;12(1):77-85.

- Battisti WP, Wager E, Baltzer L, Bridges D, Cairns A, Carswell CI, et al. Good publication practice for communicating company-sponsored medical research: GPP3. Ann Intern Med. 2015;163(6):461-4.
- International Committee of Medical Journal Editors (ICMJE). December 2017. Recommendations for the conduct, reporting, editing, and publication of scholarly work in medical journals. Available at: http://www.icmje.org/recommendations/. Accessed 03 August 2018.

# 15 PROTOCOL SIGNATURE PAGES

# 15.1 Sponsor Signature Page

| Protocol #: | VX20-445-119 | Version #: | 1.0 | Version Date: | 26 June 2020 |
|---|---|---|---|---|---|
| Study Title: A Phase 3b Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Cystic Fibrosis Subjects Ages 6 Years and Older Who Are Heterozygous for the <i>F508del</i> Mutation and a Minimal Function Mutation (F/MF) | | | | | |
| This clinical study protocol has been reviewed and approved by the sponsor. | | | | | |
| Printed Name Title | | | | | |
| Signature | _ | | Date | _ | |

# 15.2 Investigator Signature Page

| Protocol #: | VX20-445-119 | Version #: | 1.0 | Version Date: | 26 June 2020 |
|---|---|---|---|---|---|
| Study Title: A | Phase 3b Open-l | label Study Ev | aluating the Long- | term Safety and | Efficacy of |
| • | - | • | n Therapy in Cysti | • | • |
| | | | or the $F508del$ Mut | 3 | _ |
| Mutation (F/N | | , teroz j go us re | | across and a symm | |
| Widtation (17) | <del></del> | | | | |
| | | | 1.0, and agree to co | • | _ |
| | | | rning elexacaftor (H | | |
| (IVA) and this | protocol supplied | l to me by Ver | tex Pharmaceutica | ls Incorporated ( | Vertex) is |
| confidential. | | | | | |
| Printed Name | | | <del>_</del> | | |
| riinteu Name | • | | | | |
| Signature | | | | | |

#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Clinical Study Protocol Addendum for Cystic Fibrosis

Cystic Fibrosis Studies for the Following Programs

Elexacaftor/Tezacaftor/Ivacaftor (VX-445/VX-661/VX-770)

Version and Date of Protocol Addendum: Version 3.0, 29 July 2020 Replaces Version 2.0, dated 15 May 2020

> Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### **Summary of Changes to Cystic Fibrosis Clinical Study Protocols**

Vertex is currently evaluating several CFTR modulators in clinical studies for the treatment of cystic fibrosis (CF), a serious and life-threatening disease. In completed studies, treatment with these CFTR modulators has generally resulted in rapid, robust, clinically meaningful, and statistically significant improvements in clinical measures, and are generally safe and well tolerated. Adverse events (AEs) seen with these treatments are mostly consistent with common manifestations of CF disease or with common illnesses in CF subjects.

During this COVID-19 pandemic, the safety of the subjects, investigators, and site personnel participating in these clinical studies is Vertex's first priority, thus it is important to minimize any unnecessary risk to COVID-19 exposure through travel to study sites. This addendum summarizes the measures taken for ongoing CF clinical studies. These operational adjustments were implemented to align with Health Authority guidance ensuring the protection of subjects, investigators, and site personnel while maintaining compliance with GCP and minimizing impact to the integrity of the studies. Overall, the benefit-risk of these studies remains favorable.

Vertex recommends that subjects and sites refer to local guidance regarding travel restrictions. There are no operational changes to the study protocols for subjects who can travel to the study sites for their visits. However, to ensure continued safety of subjects who *cannot* travel to the study sites for their visits (for any reason due to COVID-19), specific alternative measures are being implemented to minimize the risk of exposure to COVID-19 (see table below). As the COVID-19 pandemic evolves, Vertex will continue to assess the need for additional actions to ensure the safety of all involved in these clinical studies.

Addendum Version 3.0 summarizes additional measures taken for these ongoing CF clinical studies (see table below) to ensure continued safety.

| Protocol Change | Rationale for Change | Study Number |
|---|---|---|
| Addendum Version 3.0, dated 29 July 2020 | | |
| Assessments Unscheduled visit(s) will be permissible at the discretion of the investigator(s) or Vertex. The unscheduled visit(s) may be conducted at any time during the study (including after the protocol defined last study visit) in the event assessments specified to be collected at a scheduled visit were not collected due to COVID-19. | To ensure subject safety and/or to facilitate evaluation of safety and/or efficacy if assessments are not performed per the schedule in the protocol due to COVID-19. | VX20-445-119 |
| Implementaion of measures described in addenda versions 1.0 and 2.0, as applicable. | To ensure subject safety and/or to facilitate evaluation of safety and/or efficacy while maintaining study integrity and the safety of subjects and site personnel. | VX20-445-119 |

| Protocol Change | Rationale for Change | Study Number |
|---|---|---|
| Addendum Version 2.0, dated 15 May 2020 | | |
| Addendum Version 2.0, dated 15 May 2020 Assessments Weight and height/length/stature may be assessed by subjects or their caregivers using medical grade scales and stadiometers, as indicated per protocol and per local regulation. Sites and subjects will receive training and guidance as needed on these devices. Subjects or caregivers will provide these measurements to site personnel by telephone or video call. Investigators will review results and contact subjects for follow-up as needed. All data will continue to be retained in the subject's source files. | To allow for collection of key data to assess safety and/or efficacy while maintaining study integrity and the safety of subjects and site personnel. Addendum 1 allowed for these assessments to be performed by qualified personnel conducting the in-home visits. Addendum 2 allows for these assessments to be performed by subjects or caregivers. | |

| Protocol Change | Protocol Change | Protocol Change |
|---|---|---|
| Addendum Version 1.0, dated 24 April 2020 | | |
| Consenting of Subjects ICFs may be provided electronically or by post mail to subjects (and/or caregivers, as indicated per protocol). The subjects and/or caregivers will review the ICF with an appropriately qualified member of the investigator's team via telephone contact or video call. After this review, subjects and/or caregivers will consent (or assent, if applicable), and/or reconsent verbally and by signing and dating the ICF and returning it to the site via post mail. The signed and dated ICF will then be signed and dated by the investigator. Subjects participating in select studies may have the opportunity to enroll in longterm extension studies. Informed consent (or assent, if applicable), and/or reconsent for subjects (and/or caregivers, as indicated per protocol) may be obtained per the same process described | To provide alternative methods of obtaining reconsent or consent, as applicable, while ensuring subject safety. | |
| above, as applicable. Study Drug Shipping | To ensure subjects can continue | - |
| Study drug may be shipped directly from the site to the subject, as applicable, and if permitted by local regulations; subject protected health information will not be released to Vertex. | treatment with study drug without interruption while ensuring their safety. | |
| Reconciliation, return, and destruction of study drug will continue to occur at the clinical site as indicated per protocol and in adherence to local regulations. | To clarify that despite these alternative measures, reconciliation, return, and destruction of study drug will remain as indicated per protocol. | |
| In-home Visits and/or Telephone Contact | To provide subjects the opportunity to | |
| Study visits may be conducted as in-home visits by qualified personnel as requested by participating sites on a per-subject basis. In addition, all subjects may be contacted by site personnel by telephone or video call, irrespective of in-home visits. | continue participation in the clinical<br>studies while ensuring their safety by<br>minimizing the risk to COVID-19<br>exposure through travel. | |

| Protocol Change | Protocol Change | Protocol Change |
|---|---|---|
| Addendum Version 1.0, dated 24 April 2020 | | |
| Safety Assessments and Reporting Safety assessments, as indicated per protocol, may be performed by qualified personnel conducting the in-home visits (e.g., personnel from site or qualified health care agency). These assessments may include the following, as indicated per protocol, and per local regulation: • vital signs • urinalysis • blood draws for safety test panels (chemistry, LFT panel, lipid panel, hematology, coagulation). • physical examination (complete or abbreviated) • pregnancy test (serum or urine) Blood and/or urine samples for safety assessments are analyzed as indicated per protocol for subjects who have in-home visits. | To assess the safety and tolerability of the CFTR modulator evaluated in the specific clinical study while ensuring subject safety. These safety assessments will continue to provide safety data while minimizing burden to subjects and site personnel. To clarify that despite these alternative measures, all adverse events and serious adverse events should be reported as indicated per protocol. | |
| Blood and/or urine samples for safety assessments may be collected and analyzed at local laboratories for subjects who do not have in-home visits, but do not complete the assessment at the site. | | |
| In addition, safety assessents will be evaluated by telephone. These assessments may include the review of the following: • AEs • signs and symptoms/systems for CF • medications • planned or unplanned hospitalizations for CF • study drug administration • outcomes related to PEx • outcomes related to antibiotic treatment Investigators will review results (in-home and telephone) and contact subjects for follow-up as needed. All data will continue to be retained in the subject's source files. Any clinically significant finding (e.g., AE, SAE, laboratory abnormalities) will continue to be reported as indicated per protocol. | | |

| Protocol Change | Protocol Change | Protocol Change |
|---|---|---|
| Addendum Version 1.0, dated 24 April 2020 | | |
| Efficacy and Other Assessments Efficacy and other assessments, as indicated per protocol, may be performed by qualified personnel conducting the in-home visits. These assessments may include the following, as indicated per protocol, and per local regulation. In-home Spirometry Assessment A spirometry device may be provided to subjects for in-home assessments of lung function as indicated per protocol. Sites and subjects will receive training and guidance as needed. | To be able to assess safety, treatment effectiveness, and quality of life measures of the CFTR modulator evaluated in the specific clinical study while ensuring subject safety. | |
| Patient Reported Outcome CFQ-R questionnaires may be provided to subjects (electronically or post mail) to be completed at home as indicated per protocol. Subjects will return these questionnaires to the site via post mail. | | |
| Other Assessments ECGs sweat chloride blood samples for <i>CFTR</i> genotype testing, IRT, PK, FSH, inflammatory mediator, biomarkers, and vitamin levels fecal samples for FE-1, fecal calprotectin, and other markers of intestinal inflammation other patient reported outcomes (e.g., TSQM, SF-12) | | |

| Remote Monitoring Vertex has implemented remote monitoring visits where applicable, including remote source data verification, as allowed per local regulations. Remote monitoring will focus on collection of safety data, and data supporting primary and key secondary endpoints. To allow for review of key data to inform on the safety of subjects receiving treatment. To allow for review of other key data to inform on the objectives of the study while maintaining study integrity and the safety of subjects and site personnel. | Protocol Change | Protocol Change | Protocol Change |
|---|---|---|---|
| Vertex has implemented remote monitoring visits where applicable, including remote source data verification, as allowed per local regulations. Remote monitoring will focus on collection of safety data, and data supporting primary and key secondary endpoints. To allow for review of other key data to inform on the objectives of the study while maintaining study integrity and the safety of subjects and site | Addendum Version 1.0, dated 24 April 2020 | | |
| | Remote Monitoring Vertex has implemented remote monitoring visits where applicable, including remote source data verification, as allowed per local regulations. Remote monitoring will focus on collection | inform on the safety of subjects receiving treatment. To allow for review of other key data to inform on the objectives of the study while maintaining study integrity and the safety of subjects and site | |

AE: adverse event; CF: cystic fibrosis; CFQ-R: Cystic Fibrosis Questionnaire-Revised; ECG: electrocardiogram; FE-1: fecal elastase-1; FSH: follicle-stimulating hormone; GCP: Good Clinical Practice; ICF: informed consent form; IRT: immunoreactive trypsinogen; LFT: liver function test; PEx: pulmonary exacerbation; PK: pharmacokinetic; SAE: serious adverse event; SF-12: 12-Item Short Form Health Survey; TSQM: Treatment Satisfaction Questionnaire for Medication